# Bismuth Subsalicylate's Role in the Prevention of Travelers' Diarrhea and Impact on Acquisition of Gut Antimicrobial Resistance Genes

\_\_\_\_\_

NCT: NCT03535272

Date: 12/20/23

# Table of Contents

| Project Overview | 5–9 |
|-----------------------------------------------------------------|-------|
| Protocol Summary | |
| Accelerated Protocol Review | |
| Investigators/Collaborators and Funding Mechanism | |
| Conflicts of Interest | |
| Introduction | 9–13 |
| Current State of Knowledge | |
| Justification for Study | |
| Intended Potential Use of Study Findings | |
| Study Design and Location(s) | |
| Objectives | |
| Hypotheses | |
| General Approach | |
| Procedures and Methods | 13–39 |
| Design | |
| Statement of Purpose | |
| Study Medications | |
| Procedures | |
| Duration of Subject Involvement | |
| How the Study Design Addresses the Objectives and Hypotheses | |
| Stakeholder Participation | |
| Cost Benefit/Prevention Effectiveness | |
| Description of Risks to the Participant | |
| Description of Anticipated Benefits to the Participant | |
| Description of the Potential Risks to Anticipated Benefit Ratio | |
| Emergency Care | |
| Study Timeline | |
| Study Population | |
| Description and Source of the Study Population | |
| Definitions | |

Participant Inclusion Criteria

Participant Exclusion Criteria

**Estimated Number of Participants** 

Sample Size and Power Calculation

**Recruitment and Enrollment** 

**Description and Justification of Compensation** 

Statement of Extra Costs to Participants Due to their Involvement in the Study

Procedures for Implementing and Documenting Informed Consent

Plan for Monitoring the Informed Consent Process

Variables and Interventions

Variables

**Study Instruments** 

Questionnaires

Pre-travel

During travel

Post-travel

**Laboratory Instruments** 

**Analytic Tests** 

Intervention

Outcomes

Criteria for Removal from the Study

Training for Study Personnel

Data Handling and Analysis

Data Analysis Plan

**Data Collection** 

Biologic (stool) Specimen Collection and Testing

Provision for Protecting/Privacy/Confidentiality

Information Management and Analysis Software

Data Entry, Editing and Management, and Data Storage

**Quality Control and Assurance** 

Bias in Data Collection, Measurement, and Analysis

**Study Limitations** 

Response to New or Unexpected Findings and Changes in the Study Environment

# Identifying, Managing, and Reporting Adverse Events Notifying Participants of their Individual Results Disseminating Information to the Public

| Budget Estimates | _40–41 |
|------------------|--------|
| References | _42–44 |
| Appendices | _45-75 |

APPENDIX A: Screener

APPENDIX B: Country Listing for Inclusion

APPENDIX C: Pre-travel Questionnaire

APPENDIX D: During-travel Questionnaire

APPENDIX E: Post-travel Questionnaire

APPENDIX F: Informed Consent Form

APPENDIX G: Follow-up Phone Call Schedule

**APPENDIX H: Recruitment Materials** 

APPENDIX I: Data Analysis Table Shells

APPENDIX J: Auto-Generated Email for Questionnaires

**APPENDIX K: Handout: Participant Instructions** 

# **Project Overview**

# **Protocol Summary**

The purpose of this study is to determine if the use of prophylactic bismuth subsalicylate (BSS) has an effect on the acquisition of travelers' diarrhea (TD) or antimicrobial resistance (AMR) genes in fecal samples among international travelers who departed from the United States to South East Asia, South Central Asia, or Africa. Our hypotheses will be tested using a double-blinded, placebo controlled randomized clinical trial with participants from a pre-travel health clinic in the United States (see Study Design and Location). To be eligible to participate, travelers must be at least 18 years and no older than 70 years of age, travel internationally to South East Asia, South Central Asia, North Africa, or Sub-Saharan Africa for 7 to 21 days, be non-pregnant and non-nursing, and be willing to participate. We expect, based upon prior studies (see Current State of Knowledge), to see a decreased incidence of TD among participants in the intervention group. We also believe, based upon known properties and actions of BSS, that there will be reduced acquisition of gut AMR genes in the intervention group. We hope findings from this study will be used to help international travelers prevent TD and changes to their intestinal resistome, thereby decreasing the spread of AMR genes across international borders.

#### Accelerated Protocol Review

None needed.

#### **Funding Mechanism**

This will be funded under the 28<sup>th</sup> Amendment to a Cooperative Research and Development Agreement (CRADA) between CDC and P&G (expiration: June 30, 2018). A new Amendment will be instated to allow continuation beyond the expiration date. The New York Center for Travel and Tropical Medicine clinic will be the lead of the project. Funds will also be provided directly to the New York Center for Travel and Tropical Medicine for clinic activities.

# **Investigators/Collaborators**

**Principal Investigators:** 

The New York Center for Travel and Tropical Medicine clinic director Bradley A. Connor, MD will serve as a co-Principal Investigator(s) (co-PI) with the CDC's Kristina M. Angelo, DO, MPH&TM (co-PI).

# The New York Center for Travel and Tropical Medicine:

Bradley A. Connor, MD

Clinic Director, New York Center for Travel and Tropical Medicine clinic Co-Principal Investigator

Olga Whyte, R.N.

Nurse and study personnel

Marina Rogova, R.N.

Nurse and study personnel

# **Centers for Disease Control and Prevention:**

Kristina M. Angelo, DO, MPH&TM

Division of Global Migration and Quarantine

Travelers' Health Branch

Co-Principal Investigator

# Erin Breaker

Division of Healthcare Quality Promotion

Clinical and Environmental Microbiology Branch

Jonathan Daniels, MS

Division of Healthcare Quality Promotion

Clinical and Environmental Microbiology Branch

Tom de Man, MS

Division of Healthcare Quality Promotion

Clinical and Environmental Microbiology Branch

Douglas H. Esposito, MD, MPH

Division of Global Migration and Quarantine

Travelers' Health Branch

Kirsten P. Fagerli

Division of Foodborne, Waterborne, and Environmental Diseases

Waterborne Diseases Prevention Branch

#### Cindy Friedman, MD

Division of Foodborne, Waterborne, and Environmental Diseases Enteric Diseases Epidemiology Branch

# Alison Halpin, BS, PhD

Division of Healthcare Quality Promotion

Clinical and Environmental Microbiology Branch

# Sunkyung Kim, PhD

Division of Foodborne, Waterborne, and Environmental Diseases Waterborne Diseases Prevention Branch

# Adrian Lawsin

Division of Healthcare Quality Promotion

Clinical and Environmental Microbiology Branch

# Gillian McAllister

Division of Healthcare Quality Promotion

Clinical and Environmental Microbiology Branch

# Eric Mintz, MD

Division of Foodborne, Waterborne, and Environmental Diseases Waterborne Diseases Prevention Branch

# K. Allison Perry, MS

Division of Healthcare Quality Promotion

Clinical and Environmental Microbiology Branch

# Ian Plumb, MBBS, MSc

Division of Foodborne, Waterborne, and Environmental Diseases Enteric Diseases Epidemiology Branch

# Mark Sotir, PhD

Division of Global Migration and Quarantine

Travelers' Health Branch

# Allison Taylor Walker, PhD

Division of Global Migration and Quarantine

Travelers' Health Branch

#### Nicholas Vlachos

Division of Healthcare Quality Promotion

Clinical and Environmental Microbiology Branch

Dr. Connor's team at The New York Center for Travel and Tropical Medicine will lead this study. They will perform study subject consent, enrollment, double-blinded assignment of study subjects to intervention and placebo groups, data (both questionnaires and biologic [stool] sample) collection, and response to traveler questions during travel as required. They will also manage the IRB submission.

Dr. Angelo's team in the Travelers' Health Branch at CDC will assist with the study design and protocol development, conduct the blinding of placebo and intervention medications, perform data analysis of both questionnaire and biologic (stool) specimen data including data interpretation (with coded data), and provide epidemiologic and travelers' health subject matter expertise and support to Dr. Connor's team.

Any publications using this data will require with the New York Center for Travel and Tropical Medicine clinic's involvement and oversight. CDC will not interact with any research subjects or have access to or handle any personally identifiable information, with the exception of a limited number of information technology personnel responsible for REDCap software maintenance, who are not participating in the study or protocol. CDC will not retain or claim ownership of the resulting data. CDC will be providing a secure data management platform (REDCap) to the New York Center for Travel and Tropical Medicine; CDC will have access to de-identified data only with the approval of Dr. Connor and his team. A nondisclosure agreement with The New York Center for Travel and Tropical Medicine will be signed; the clinic will not provide any PII (or the key to the coded PII) to any CDC staff.

The Clinical and Environmental Microbiology Branch at CDC will assist with study design, receive all biologic (stool) specimens for testing (coded; no PII will be sent with the specimens), and perform all laboratory analyses as indicated per the protocol. They will also store biologic (stool) specimens for further analysis.

The Enteric Diseases Epidemiology Branch at CDC will assist with study design and protocol development, data interpretation, and will provide epidemiological, statistical, and enteric diseases subject matter expertise and support.

P&G will not be involved with execution of the protocol. They will provide all intervention and placebo group medications and funding for the study.

#### **Conflicts of Interest**

P&G states that their purpose is to improve the lives of the world's consumers, and are interested in knowing whether their products and services are effective in this capacity. Because it is a publicly-traded private, for-profit corporation, P&G must develop products that consumers find useful enough to purchase regularly. This study will help the company understand more fully how its products further their mission to improve lives, may help the company develop new marketing strategies for their products, or modify existing formulations of their products to be more effective at preventing intestinal colonization with potentially harmful microorganisms.

# Introduction

# **Current State of Knowledge**

Travelers' diarrhea (TD) is the most common travel-related illness reported by international travelers, affecting between 30-70% of all travelers (1). The incidence of TD varies by travel destination, duration of travel, season, travel activities, and personal traveler attributes. Some areas of the world are considered high-risk, including Asia and Africa, but also the Middle East, Mexico, and Central and South America (1). Previous placebo-controlled clinical trials with the prophylactic use of bismuth subsalicylate (BSS) demonstrated a significant reduction in the incidence of TD among those receiving the drug. A recent unpublished meta-analysis on the subject of BSS prophylaxis found that persons who took BSS while traveling internationally before the onset of gastrointestinal symptoms had a 3.5 times greater odds of remaining free of TD in comparison to those who received placebo (2). BSS is available in both liquid and tablet formulations; both formulations reduced TD at doses of either 60mL four times daily (4.2g/d) for the liquid formulation (3) or 2 tablets, four times daily (2.1 g/day) for a maximum of 3 weeks (3, 4, 5). BSS at 2.1 g/day protected 41–65% of participants (3, 5), while the liquid formulation protected 62% of participants (3). Studies suggest the lowest minimum dose for protection may be 1g daily taken in 2 doses, which provided 35% protection in one analysis (5) and 40% protection in others (3, 4). BSS had minimal side effects, but these may include nausea,

constipation, tinnitus, and blackening of the tongue and stool (5, 6). BSS may cause encephalopathy if taken in high doses for prolonged periods, but this is exceedingly rare and above the recommended dose (7, 8).

The active component of BSS with antimicrobial effects is bismuth, which is poorly absorbed and mostly remains in the GI tract while salicylate is systemically absorbed in the stomach (9). The mechanism of action of BSS in the prevention of TD is thought to be due to bismuth's intraluminal antimicrobial properties and a reduction in the number of bacteria (4, 6, 9, 10). Invitro studies suggest that bismuth's action is bactericidal (6, 11), even at various levels of intestinal pH and against a wide range of organisms (11). The precise mechanisms of action include the binding of ingested bacteria and subsequent marking of these organisms to be killed by host defenses, rendering the bacteria unable to attach to receptor sites that are important for colonization and infection (11), degrading the bacterial cell wall, inhibiting ATP synthesis, and inhibiting the function of the plasma membrane (9). This inhibition may occur in as little as 0.5–24 hours (9). BSS may also inactivate bacterial toxins before attachment to the intestinal mucosa (12). Viruses may be inhibited by BSS; it may prevent viral invasion and deter replication through unknown mechanisms (4).

There is a current domestic and international focus on preventing the acquisition of drugresistant enteric bacteria by high-risk groups, including travelers (13). International travelers are at increased risk for acquiring gut organisms containing AMR genes (especially after travel to Asia), developing TD, taking antibiotics, and requiring hospitalization (14, 15, 16, 17). Although carriage of organisms containing gut AMR genes may be transient in most travelers (15), it can persist for ≥1 year in over 10% of travelers, increasing the risk of transmission to household members and others (18). Avoiding the use of antibiotics while abroad is one way to lessen acquisition of antibiotic-resistant organisms (19). BSS treatment of adult outpatients with acute diarrhea has been found to reduce antimicrobial medication use in a high prevalence area (20). It is currently unknown whether BSS affects the acquisition of gut AMR genes while traveling abroad; however, given BSS' antimicrobial properties, stability in acidic conditions, and blockage of receptor sites to prevent colonization, it is possible that prophylactic BSS may indirectly prevent acquisition of AMR genes in international travelers by preventing intestinal colonization of ingested microbes. More research must be done to address this uncertainty.

# **Justification for Study**

International travel has expanded over the past 50 years. Worldwide annual tourist arrivals are expected to reach 1.8 billion by 2030 (21). Travel destinations continue to diversify, including increasing numbers of travelers visiting countries with emerging economies, such as Asia and Africa. These trends may place international travelers into closer contact with infectious pathogens, including those that cause TD and have AMR genes (21, 22). This may contribute to infectious disease spread across international borders. International travel, particularly to countries with emerging economies, is a well-documented risk factor for acquisition of gut AMR genes (23, 24). Also, acquisition of TD during travel has been associated with persistent infection or post-infectious irritable bowel syndrome (PI-IBS). PI-IBS is the onset of irritable bowel symptoms after an enteric infection, and may lead to a permanent change in bowel function (25).

Given the burden of TD and the possibility of acquiring AMR genes while abroad, there is ample justification for studying simple, cost-effective, and safe actions that could be taken by international travelers to reduce these risks.

#### **Intended Potential Use of Study Findings**

Healthcare providers and public health officials may use the findings from this study to enhance or change recommendations made to international travelers when offering pre-travel advice. Healthcare providers may advise travelers on improved best practices to decrease their risk of TD and acquisition of AMR genes. Public health officials may use information from this study to develop guidelines and advise on best practices to ensure that the impact of TD and drugresistant organisms is minimized in international travelers. By minimizing acquisition of AMR genes in international travelers, we would also be helping protect the general, non-traveling public from exposure to imported antimicrobial resistant organisms. This study may also generate hypotheses that could help guide future study of possible mechanisms of action and uses of BSS in reducing the development of and treating TD.

The results will be made public through publication(s) within 18 months of the termination of data collection. This/these publication(s) will be in a peer-reviewed journal; however, the initial release may be in the form of an abstract and presentation at a scientific meeting (see Disseminating Information to the Public).

# Study Design and Location(s)

This study will be conducted as a double-blinded, placebo-controlled randomized clinical trial. We propose two arms to test BSS against placebo:

- 1. BSS 4 tablets po bid (2.1 grams total of BSS)
- 2. Placebo 4 tablets po bid

Study participants will be recruited from The New York Center for Travel and Tropical Medicine Clinic in New York, New York, USA (see Procedures) (<a href="http://www.travelhealth.net/">http://www.travelhealth.net/</a>). Throughout the study period, the recruiting site will maintain adequate personnel trained in the study protocol and procedures (see Training for Study Personnel). Study personnel will be available to communicate with the co-PIs as necessary and to address issues with the study protocol and concerns of the study participants. This site will be able to consent and enroll participants (see Procedures for Implementing and Documenting Informed Consent), store and distribute the study drug and placebo, and collect and safely store questionnaire data (see Data Handling and Analysis) and biologic samples (stool) data (see Biologic [stool] Specimen Collection and Testing), in accordance with the study protocol.

#### **Objectives**

- 1. (Hereafter, "primary objective") Test the efficacy of BSS in the prevention of TD among international travelers.
- 2. (Hereafter, "secondary objective") Determine the impact BSS has in the acquisition of gut AMR genes among international travelers.

# **Hypotheses**

The following hypotheses follow the objectives above:

- 1. NULL HYPOTHESIS: BSS does not prevent TD among international travelers.
  - a. Does BSS prevent TD among international travelers?
  - b. Does BSS reduce severity/frequency of TD among international travelers?
- 2. NULL HYPOTHESIS: BSS does not alter the acquisition of gut AMR genes among international travelers.
  - a. Does BSS affect the acquisition of gut AMR genes among international travelers?

- b. Does BSS affect the acquisition of gut AMR genes among international travelers that develop TD?
  - i. Does BSS alter the acquisition of gut AMR genes if an international traveler with TD takes an antimicrobial while taking BSS?
- c. Does BSS affect the acquisition of gut AMR genes among international travelers that do not develop TD?

# **General Approach**

The approach of this study will be hypothesis-testing.

#### **Procedures and Methods**

# Design

#### Statement of Purpose

The purpose of this study is to investigate the impact of BSS on the acquisition of TD and acquisition of gut AMR genes among international travelers.

# **Study Medications**

The placebo, produced by P&G, will be comprised of the following components: microcrystal cellulose, calcium carbonate, D&C red No. 27 aluminum lake, flavor, magnesium stearate, mannitol, povidone, saccharin sodium, and talc. It will be formulated to have an appearance (size, shape, color, and packaging), texture, and taste similar to BSS.

Each bottle to be used in the study will be blinded by CDC personnel (but not the co-PI). Each bottle will include an internal study ID#, owner name, batch number, start date, and expiration date. The blinding label will additionally include a study ID for identification. Bottles of study medications will be sent to The New York Center for Travel and Tropical Medicine clinic for distribution to participants at their pre-travel consultation/enrollment visit.

#### Procedures

This study will be in the form of a double-blinded, placebo-controlled randomized clinical trial, conducted at The New York Center for Travel and Tropical Medicine clinic in

New York (see Description and Source of the Study Population). This clinic offers pretravel specialty medical services to persons planning international travel and has the necessary resources, skills, and expertise to evaluate and treat travelers who acquire travel-related illness, and offer advice to travelers when questions or problems arise during their trips.

All travelers who are seen for a pre-travel consultation at The New York Center for Travel and Tropical Medicine will be administered the screening questionnaire by study personnel upon arrival to their consultation to determine their eligibility. Eligible travelers will be invited to participate in the study (see Participant Inclusion / Exclusion Criteria). All participants will be consented as per the protocol (see Procedures for Implementing and Documenting Informed Consent). Randomization of participants will be double-blinded and conducted via block randomization to ensure groups of equal sample sizes using a computer generated distribution. Study medications for both the intervention and placebo group will be provided by P&G, blinded by CDC (using a unique identifier), and distributed to participants at the clinic site during the pre-travel consultation/enrollment visit per the randomization mentioned above (see Study Medications). Study personnel at The New York Center for Travel and Tropical Medicine will not be aware of which medications are BSS or placebo. The code number of the medication (intervention or placebo) administered to a particular participant will be recorded. All code numbers and corresponding arms will be kept secret until the end of the trial.

Web-based questionnaires will be administered during and post-travel (see Study Instruments). Pre-travel data will be collected via telephone with study personnel. Pre-travel data will include information on the participant's medical history and travel plans, and post-travel data will include information on the TD symptoms, medication use, medical care received, and adverse events. During travel, the participant will complete a daily questionnaire that will include data on compliance with taking the study tablets, presence of symptoms of TD, onset of adverse reactions, any medical care received, and trip specifics. The during-travel questionnaire will be made available in both a web-based electronic form and a paper form in the event that the participant does not have reliable internet access. Any paper forms that were completed will be returned by mail

after they return from travel via a pre-paid envelope addressed to the study clinic that was given to the participant when enrolled.

To address the secondary objective, participants will also be asked to provide pre- and post-travel biologic (stool) samples for laboratory testing for the presence of gut AMR genes (see Laboratory instruments). Timing of the pre- and post-travel data and stool sample collections will be within 7 days before departure and 10 days after return from travel, respectively. Both biologic (stool) samples will be self-collected and submitted by mail to the clinic (the collection kit, and all necessary packaging and postage will be provided to the traveler). The participant will not be seen by a healthcare provider involved with the study post-travel unless they are ill and seek an evaluation.

As part of standard pre-travel consultation practices, if indicated, travelers will be prescribed anti-diarrheal medications and/or antibiotics for self-treatment of TD. These medications may include loperamide (Imodium), diphenoxylate and atropine (Lomotil), BSS (Pepto bismol), ciprofloxacin, azithromycin, or rifaximin. If these medications are taken while abroad, the travelers will be asked to note this on the during travel or post-travel questionnaires.

No difference in pre-travel advice, provision of anti-diarrheal medications, or during- or after-travel medical evaluation or advice will occur based on the traveler's assigned study arm.

#### **Duration of Subject Involvement**

The duration of each participant's involvement in the study is expected to be a maximum of 6 weeks. This will account for time to complete the pre-travel consultation/enrollment visit, 21 days (or less) of travel, and post-travel follow-up.

#### How the Study Design Addresses the Objectives and Hypotheses

A double-blinded, placebo-controlled randomized clinical trial is the best study design to address the study objectives and hypotheses. We aim to determine if there is a biologic benefit to an intervention (BSS administration), and a placebo-controlled methodology is required to determine if there is a statistically significant benefit of the intervention

regarding incidence of TD and acquisition of gut AMR genes. It is imperative to blind both healthcare providers and participants to ensure that biases, including selection and observer bias, are minimized.

#### Stakeholder Participation

The primary stakeholders for the project are international travelers, healthcare providers, and public health officials.

P&G cannot participate in the study procedures (i.e., data collection or analysis) to minimize the potential for any commercial influences or the appearance thereof. They will not be able to prevent the publication of negative results, nor influence the interpretation of the results. They will be responsible for providing both intervention medication and placebo.

CDC and P&G will operate under the terms of the CRADA regarding cooperative research, reports, financial and staffing obligations, patent applications, licensing, proprietary rights and publication, representations and warranties, disputes, and liability.

# **Cost Benefit/Prevention Effectiveness**

A single 262mg tablet of BSS costs approximately \$0.26 when purchased over-the-counter (\$10.49 for 40 tablets). The cost of antibiotic treatment of TD or potential hospitalization from complications, or for diagnostic procedures or other treatment interventions, far surpasses the cost of BSS for possible TD prevention.

The cost benefit regarding the secondary objective is unable to be defined, however, the potential costs for spread of gut AMR genes from colonized international travelers are presumed to be large compared to the minimal cost of BSS prophylaxis. Further, there is no evidence currently that any microbial resistance to BSS exists, inducible or otherwise. Finally, any reductions in TD incidence among travelers that is related to prophylactic BSS use could result in a reduced need for and use of antibiotics by travelers, with a concomitant reduction in the selective pressures for antimicrobial resistance genes.

#### Description of Risks to the Participant

There are minimal risks to participants in this study. BSS has been marketed in the United States for over 100 years, and is widely available without a prescription. It has a good safety profile at the recommended dose and duration of use. We will not exceed these safe dosing ranges in this study. The maximum daily dose (4.2g per day) of BSS results in peak serum concentrations of salicylate considerably below toxicity levels. This dose has been documented to be safely used for up to 3–4 weeks (26). We will include only adult participants and exclude children <18 years of age or elderly adults 70 years of age or older, pregnant or breastfeeding women, participants with a known contraindication to BSS use, or anyone taking medications known to interact with BSS, including other salicylate-containing compounds. Participants will be asked to refrain from taking aspirin or aspirin-containing compounds. The duration of BSS administration in this study will be limited to a maximum of 21 days.

BSS lists possible side effects on its packaging (including, but not limited to, constipation and tinnitus) that will all be discussed with the participant before informed consent and enrollment.

Participants will be provided contact information for study personnel at The New York Center for Travel and Tropical Medicine in the event that they have questions regarding the study or the medications before, during, or after travel. They will be notified to contact study personnel at The New York Center for Travel and Tropical Medicine in the event that they experience any adverse events of BSS or symptoms of TD.

In addition to the study preparations (BSS or placebo tablets), participants may also be provided with an appropriate medication for TD self-treatment (at the discretion of the healthcare provider) to carry with them in the event they develop TD while abroad. If they experience an episode of TD, they will be instructed to continue their study medication. Participants will also be counseled on hydration, the indications for antibiotic use (*i.e.*, in the event of severe diarrhea, but not mild or moderate diarrhea), and when to seek healthcare.

Each participant's confidentiality will be rigorously maintained (see Procedures for Implementing and Documenting Informed Consent). If a breech occurs, the IRB will be notified immediately and standard procedures will be followed.

#### Description of Anticipated Benefits to the Participant

Based upon published reports, we anticipate that participants in the intervention arm of the study will experience a health benefit; they will be less likely to acquire TD while abroad. They also may benefit, in the event that they do acquire TD, by having a shorter duration and lesser severity of TD symptoms in comparison to those in the placebo group.

# <u>Description of the Potential Risks to Anticipated Benefit Ratio</u>

The potential benefits of participating in this study outweigh the minimal risks.

# **Emergency Care**

We do not anticipate participants needing emergency care as a part of this study. Participants will be provided phone and email contact information for study personnel in the event questions or concerns arise that may relate to their participation in the study.

#### **Study Timeline**

Table 1. Study Timeline, 2017-2020

| Study Component | Date of Anticipated Start | Date of Anticipated End |
|---|---|---|
| Protocol Writing and Coordination | March 2017 | October 2017 |
| Submission of protocol/consent forms | November 2017 | Late December 2017 |
| for IRB approval | | |
| Training of study personnel | January 2018 | January 2018 |
| Enrollment of participants | February 2018 | July 2019 |
| Laboratory analysis of stool specimens | February 2018 | October 2019 |
| Data entry | February 2018 | October 2019 |
| Data analysis (every 3 months) | April 2018 | November 2019 |
| Manuscript writing and clearance | November 2019 | March 2020 |
| Dissemination of findings | March 2020 | |

# **Study Population**

# Description and Source of the Study Population

Participants will be selected from persons seeking a pre-travel consultation at The New York Center for Travel and Tropical Medicine, New York, United States. This clinic serves travelers by providing pre-travel consultative services, in addition to post-travel screening, assessment, diagnostic, and treatment services. Centrally located in Manhattan, this clinic serves a large variety of international travelers, including tourists, immigrants or their relatives, and business travelers, among others. Travelers' destinations are equally varied, reflecting the ethnic and cultural diversity of New York City.

# **Definitions**

#### Diarrhea:

≥ 3 unformed stools in 24 hours, with or without associated symptoms such as fever, cramping, or abdominal pain

#### Travelers' diarrhea:

Diarrhea that begins while traveling (after arrival in a country) or within 10 days after return

# Study period:

Includes the 7 days prior to departure in which the pre-travel questionnaire and a biologic (stool) specimen is collected, the full duration of travel, and through 10 days maximum post-return from travel, or until both the post-travel questionnaire and submission of the post-travel biologic (stool) specimen is complete (a maximum of 17 days post-travel)

#### Travel companion (group):

Two or more study participants with a common relation (friends, colleagues, or relatives) with the same itinerary, who anticipate performing the same activities during travel

#### Trip duration:

The number of days spent in country; excludes air travel time

#### Severe TD:

Hospitalization to an inpatient ward either during travel or after travel with a diagnosis of diarrhea

# Acquisition of AMR gene(s):

The presence in a post-travel biologic (stool) specimen of one or more antimicrobial resistance gene(s) that were not present in a pre-travel biologic (stool) specimen from the same person, and which is known to confer antimicrobial resistance to one or more antimicrobial agents ("resistome")

# Medication compliance:

Full = participant takes all scheduled doses according to directions Good = If < 15% of BSS or placebo doses were missed during travel Fair = If 15-30% of BSS or placebo doses were missed during travel Poor = If > 30% of doses were missed during travel

# Questionnaire compliance:

Full = participant completes all questionnaires

Good = participant completes >80% of all during travel questionnaires, AND both the pre- and post-travel questionnaires

Fair = participant completes between 30–80% of all during travel questionnaires, including AT LEAST the pre-travel questionnaire

Poor = participant completes <40% of all during travel questionnaires, and AT LEAST the pre-travel questionnaire

#### Biologic (stool) specimen compliance:

Full = BOTH specimens collected and sent

Fair = ONLY one specimen collected and sent

Poor = No specimens collected and sent

# Loss to follow-up:

Failure to complete the post-travel questionnaire after three attempts to contact the participant or if submission of the post-travel biologic specimen (stool) occurs more than 10 days after return from travel or is not submitted

# Participant Inclusion Criteria

Willing participants must meet the inclusion criteria as outlined here:

- 1. Be  $\geq$  18 and <70 years of age at the time of enrollment
- Sign an informed consent (see Procedures for Implementing and Documenting Informed Consent) stating willingness to participate and comply with the study protocol
- 3. Plan on leaving for an international trip ≥7 days after their pre-travel consultation
- Plan on traveling in country for ≥7 days but ≤21 days (21 day limit due to BSS duration recommendations and a lack of data on longer-term BSS use) (see
  Definitions)
- 5. Traveling to either South East Asia, South Central Asia, North Africa, or Sub-Saharan Africa for at least 7 days of their itinerary (see **APPENDIX B** for list of countries classified to each region)
- 6. Be willing to complete an initial eligibility screening (see Recruitment and Enrollment)
- 7. Be willing to complete questionnaires and provide biologic specimens (stool) within 7 days of departure and within 10 days after return
- 8. Be willing to refrain from taking any pre-biotics, probiotics, synbiotics and/or herbal supplements throughout their study period

# Participant Exclusion Criteria

Willing participants must not meet any exclusion criteria as outlined here:

- 1. Are <18 years of age or >69 years of age
- 2. Are traveling in country for <7 or >21 days (see Definitions)
- 3. Have known or suspected contraindications to taking BSS (including, but not limited to, travelers with kidney disease, diabetes, gout, a clotting disorder, or an allergy to any component of BSS)

- Are pregnant (via self-report), are planning to become pregnant, or may become
  pregnant during travel (not actively using contraception and are sexually active), or
  are breastfeeding
- 5. Routinely take a medication known to interact with BSS (including, but not limited to, insulin, methotrexate, valproic acid, ACE inhibitors, anticoagulants, or other salicylates) (see **APPENDIX A** for complete list)
- 6. Have taken an antibiotic in the 30 days before departure
- 7. Have taken any medications that may lower one's ability to fight infection (e.g., steroids, monoclonal antibodies, etc.)
- 8. Have previous diagnoses of immunocompromising conditions such as HIV/AIDS, complement deficiency, immunoglobulin deficiency, or undergoing active chemotherapy or participants with chronic gastrointestinal disorders, such as chronic diarrhea, irritable bowel syndrome (IBS), inflammatory bowel disease (i.e., Crohn's disease, ulcerative colitis), celiac disease, malabsorption syndromes, pancreatic insufficiency, gallbladder disease, or current gastrointestinal cancer
- 9. Have had diarrhea (see Definitions) anytime in the previous 30 days, have diarrhea at the pre-travel consultation, or develop diarrhea before departure
- Have been given doxycycline for malaria prophylaxis for the current trip (due to possible drug-drug interactions and decreased absorption of the doxycycline) (27)
- 11. Have an allergy to any component of the placebo tablets

# **Estimated Number of Participants**

We anticipate enrolling approximately 500 participants (see Sample Size and Power Calculation).

# Sample Size and Power Calculation

A sample size of 488 participants with full compliance to medications and questionnaires (244 participants in each arm) is needed to fulfill the objectives [anticipated incidence of the endpoint as 40% incidence of TD with a 30% minimum intervention protection (0.40-[0.4x0.30]= 0.28) with an alpha of 0.05, and 80% power].

# Recruitment and Enrollment

All international travelers undergo a screening questionnaire at their pre-travel consultation to determine eligibility. This short questionnaire includes questions regarding the travelers' [see **APPENDIX A**]:

- 1. Age
- 2. Travel destination(s)
- 3. Trip duration
- 4. Acute and chronic medical conditions, including diarrhea
- 5. Contraindications to BSS administration
- 6. All current medications, including antibiotic use within the 30 days before screening
- 7. Willingness to participate in the trial and comply with the data collection requirements

This screening questionnaire will be administered to the traveler by study personnel at The New York Center for Travel and Tropical Medicine. The purpose will be to exclude those travelers who do not meet all inclusion criteria and those who meet any exclusion criteria (see Participant Inclusion / Exclusion Criteria). Travelers who meet the inclusion criteria and do not meet any exclusion criteria will be introduced to the project objectives and procedures, including the procedures for biologic (stool) specimen collection (see Laboratory instruments).

Once recruited and consented, eligible participants will be registered in the study at the clinic site and receive a one-page instructional handout regarding stool specimen collection and questionnaire completion [APPENDIX K]. All primary participant information will be kept at the clinic. Travelers will agree to inform the study personnel at their clinic site if they have a change in travel plans, begin a course of antibiotics, become pregnant before or during travel, or develop diarrhea before departure, to determine if they are still eligible to participate. In the event that a participant withdraws from the study at any time, the clinic must note this in the study database.

#### Description and Justification of Compensation

Gift card compensation will be provided to the participants for the time spent on this project.

The participant will receive \$100 for completion of the pre-travel questionnaire and the submission of a pre-travel biologic (stool) specimen. For each daily questionnaire that the participant completes while traveling, they will receive an additional \$5 (maximum additional \$100). The participant will receive an additional \$50 for completion of the web-based post-travel questionnaire and an additional \$50 for the submission of a biologic (stool) specimen post-travel. The maximum compensation will be \$300 total. The minimum participation to receive compensation is good medication compliance, good questionnaire compliance, and good biologic (stool) specimen compliance (see Definitions).

Compensation will be mailed to participants upon completion of their study period.

# Statement of Extra Costs to Participants Due to their Involvement in the Study

We do not anticipate any extra costs to the participants due to their involvement.

# Procedures for Implementing and Documenting Informed Consent

The New York Center for Travel and Tropical Medicine clinic must obtain and ensure scientific and ethical permission, in accordance with state and national regulations. All collaborators must adhere to strict guidelines to ensure participant confidentiality, following the Privacy Act. Biological specimens (stool) must be processed per established safety protocols.

Each participant will provide written informed consent for the project at their initial pretravel consultation when they are enrolled by study personnel (see **APPENDIX F**). This will include (but is not limited to) information regarding the study objectives and rationale, the study procedures, how each participant's confidentiality will be protected, their rights as participants, and compensation for participation. It will also include information on how their biologic specimens will and will not be used. Study personnel will answer the travelers' questions pertaining to study logistics and BSS as necessary.

Participants may withdraw from the study at any time. Participants will self-monitor for BSS side effects and the study will be suspended in the event of safety concerns.

#### Plan for Monitoring the Informed Consent Process

Each informed consent will be signed in the presence of a witness to ensure all risks and benefits, in addition to an explanation of confidentiality, were described to the participant.

#### **Variables and Interventions**

#### Variables

Variables collected on participants are available in the **APPENDICES**. They are also described in further detail below.

# **Study Instruments**

Questionnaires (see APPENDICES)

Any revisions to study procedures or instruments will be submitted to the IRB as an amendment for approval before changes are implemented.

#### Screening (see APPENDIX A)

# Pre-travel (see APPENDIX C)

Contact information (phone and email) for each participant who consented at the pre-travel consultation/enrollment visit will be given to the study personnel who will administer the screening questionnaire. Each participant will be contacted via telephone 7 days before departure, and study personnel will review the participant's responses to each question on the screening questionnaire to ensure they are still eligible to participate. At this time, they will complete the pre-travel questionnaire with the participant on the phone and answer any questions they may have. The participant will also be reminded to submit their pre-travel biologic (stool) specimen.

Study personnel will make follow-up telephone calls on pre-departure days 7, 5, 3, and 1 as needed to ensure the questionnaire is completed.

This questionnaire will include information from the eligibility screening, in addition to the following information:

- 1. Demographics (e.g., age, sex, and ethnicity)
- 2. Medical history
- Current medications (including use of probiotics, over-the-counter medications, or herbal supplements)
- 4. Previous international travel in the past 90 days
- 5. Travel plans including destination(s) and duration
- 6. Reason(s) for travel

# During Travel (see APPENDIX D)

During travel, participants complete a daily questionnaire that will include the following information:

- Date, time, and number of study tablets taken (to provide information on the number of missed doses)
- 2. Presence of gastrointestinal symptoms (e.g., abdominal cramping, fever, nausea, vomiting, tenesmus)
- 3. Duration of GI symptoms
- 4. Possible medication adverse reactions (e.g., tinnitus, black stool, etc.)
- 5. Other illnesses acquired (e.g., upper respiratory infection)
- Hospital admission or contact with a healthcare facilities or providers or taking any non-routine medications for illness while abroad
- 7. Countries visited
- 8. Foods eaten (fermented foods or yogurt)

Details on the participant's trip (number 7 above) are necessary to determine risk factors for the acquisition of gut AMR genes among those participants in the placebo group vs the intervention group.

Web-based data collection will be used to facilitate data collection during travel. Each participant will receive a unique URL to input their

daily information using their unique Study ID and Group ID. A paper copy of the daily travel questionnaire will be provided as a back-up mechanism for data capture where internet access is limited or unavailable. If a participant does not think that they will have reliable internet access while abroad, they will be encouraged to use the paper copies to ensure real-time data collection. Labels will be provided to ensure that the paper copies are de-identified. Any paper forms that were completed will be returned by mail after they return from travel via a pre-paid envelope addressed to the study clinic that was given to the participant when enrolled (see Procedures).

Participants will take either BSS or placebo for the duration of travel, unless they reach a study outcome or criteria for removal (see Outcomes and Criteria for Removal from the Study).

# Post-travel (see APPENDIX E)

Participants will be asked to submit a web-based post-travel questionnaire within 10 days after return from travel, submit a biologic (stool) specimen, and provide all daily questionnaires that were completed during travel. This will be submitted via a pre-paid envelope addressed to the study clinic that was given to the participant when enrolled.

Study personnel will make follow-up telephone calls on days 3, 5, 7, and 10 after return as needed to encourage that the post-travel questionnaire, paper questionnaires from during-travel, and biologic (stool) specimens are all submitted.

The web-based post-travel questionnaire will include questions on:

- The development of symptoms of TD since returning from abroad, including duration of symptoms
- 2. New antibiotic or other medication use
- 3. Adverse events

- 4. Contact with healthcare facilities or providers
- 5. Changes to travel itinerary during travel

Table 2. Schedule of CLINIC events (primary and secondary objectives):

| | Stages | | | |
|---|---|---|---|---|
| | Pre-travel | Pre-travel | During | Post-travel |
| | consultation | (≤7 days | travel | (≤10 days |
| | (baseline) | before | | after return) |
| | | departure) | | |
| Screening Questionnaire | Х | | | |
| Informed Consent | Х | | | |
| Pre-travel | | Х | | |
| Questionnaire* | | | | |
| Follow-up call(s) | | Х | | X <sup>†</sup> |
| During travel | | | Х | |
| Questionnaires | | | | |
| Post-travel | | | | Х |
| Questionnaire | | | | |
| Adverse Events Reporting | | | Х | Х |

\*Study personnel will call the participant to complete a pre-travel questionnaire 7 days before departure and to ensure that answers to the questions on the screening questionnaire have not changed. Reminder calls will occur as per **APPENDIX G**. If the traveler is leaving exactly 7 days after the pre-travel consultation/enrollment visit, this questionnaire can be performed at the pre-travel consultation/enrollment visit.

<sup>†</sup>Study personnel will call the participant within 3 days of return from travel to remind participants to complete their web-based post-travel questionnaire, submit any paper during travel questionnaires, and collect and submit the post-travel biologic (stool) sample. Reminder calls will occur as per **APPENDIX G.** 

# **Laboratory Instruments**

All participants will collect and submit a fresh biologic (stool) sample in the 7 days before departure and within 10 days after return. Participants will be

provided all instructions and materials necessary to collect and submit these samples at enrollment. All biologic (stool) specimens will be submitted by mail, and participants will be given pre-paid shipping materials.

Participants will be provided two OMNIgene gut kits at their pre-travel consultation/enrollment visit once enrolled (see Biologic [Stool] Specimen Data Collection and Testing). These kits will come with instructions on use, handling, and shipment.

In the event that participants are able to provide a stool sample while in clinic for their pre-travel consultation/enrollment visit or during a non-study post-travel follow-up sick visit within 10 days of return, these samples will be aliquoted by study personnel at The New York Center for Travel and Tropical Medicine in the following manner:

\*First, the required quantity will be placed in the participant's OMNIgene gut kit (per manufacturer directions) to be sent to CDC's Clinical and Environmental Microbiology Branch for resistome testing. The remainder will be frozen, and sent to CDC for analysis at a later date (note: OMNIgene gut kit does not allow for culture - a see Biologic [Stool] Specimen Collection and Testing). Only those participants who happen to have a biologic (stool) specimen collection completed at the clinic will have their stool analyzed by culture; this is not a requirement for participation and no additional compensation above that previously described will be offered.

Table 3. Schedule of LABORATORY events (secondary objective)
(Events from Table 2 still apply to these participants)

| | Stages | | |
|-----------------------------|------------|---------------|-------------|
| | Pre-travel | During travel | Post-travel |
| Biologic (stool) sample | X | | Х |
| Laboratory testing of stool | Х | | Х |

Analytic tests

Questionnaires: Data from the questionnaires will be analyzed for statistical significance comparing intervention vs placebo groups.

Biologic (stool) specimens: A highly multiplexed PCR assay detecting over 500 different AMR genes will be used to test the DNA extracted from all biologic (stool) specimens that were placed in the OMNIgene gut kit (see Biologic (Stool) Specimen Collection and Testing). Results will be analyzed to determine if the participants acquire gut AMR genes (changes to the "resistome") as a result of travel and whether or not that change varied with the bismuth subsalicylate treatment received. Additionally, stool bacteriologic culture will be performed on those specimens submitted in clinic.

#### **Intervention**

We propose the inclusion of two arms to test BSS against placebo:

- 1. BSS 4 tablets po bid (2.1 grams total)
- 2. Placebo 4 tablets po bid

Dosing will begin on the flight prior to arrival in the destination and will cease once they return home. The study medications must be taken twice daily (a morning and an evening dose); with time zone changes, the first dose should be taken to ensure that no longer than 12 hours passes before a subsequent dose.

Before departure, participants will be provided, free of charge, all needed study medication for the duration of their trip. Participants will be encouraged to take all doses of their medication and appropriately document on their daily during travel questionnaires if a dose was missed or taken off schedule.

# **Outcomes**

The outcomes of this study will include:

| | Favorable Outcome | Non-favorable Outcome |
|---|---|---|
| Hypothesis 1: | Prevention of TD in the | TD in the intervention group at a |
| Prevention of TD | intervention group | rate similar to placebo; intervention |
| | | drug side effects; adverse events |

| Hypothesis 2: | Reduced or no presence of | No reduction in the presence of |
|---|---|---|
| Acquisition of AMR | travel-associated gut AMR | travel-associated gut AMR genes in |
| genes | genes in the intervention | the intervention group |
| | group | |

The participant's study period will end in the following circumstances:

- 1. The traveler meets criteria for removal (see Criteria for Removal from the Study)
- 2. The participant voluntarily withdraws from the study (see Procedures for Implementing and Documenting Informed Consent)
- 3. The participant completes all study activities and submits all study questionnaires and biologic (stool) specimens
- 4. The participant is lost to follow-up

The participants will be instructed at enrollment to stop the study medication for any of the following reasons (although they will still be instructed to answer their questionnaires and submit biologic [stool] specimens as scheduled):

- Antibiotics or BSS (either provided by the study personnel for TD treatment, or taken as an over-the-counter remedy) are taken for TD or for another medical condition
- 2. Any severe adverse events as described, such as signs and symptoms of salicylism or neurotoxicity, occur
- 3. Hospitalization for any reason

Barring the reasons listed above, the study medication should be taken throughout the trip duration, even if diarrhea occurs, if possible.

#### Criteria for Removal from the Study

Participants will be removed from the study when any of the following criteria apply:

- 1. Do not complete the pre-travel questionnaire (see Definitions for compliance)
- 2. Loss to follow-up (see Definitions)
- 3. Voluntary withdrawal of consent by the participant for any purpose at any time
- 4. Pregnancy
- 5. Death

6. Co-PIs decide to remove a participant because of safety or integrity of the study

In the event of removal for reason #6 above, participants will still be compensated for their participation in the study (see Description and Justification of Compensation).

The date and reason for removal will be documented in the study records.

# **Training for Study Personnel**

All study personnel at the The New York Center for Travel and Tropical Medicine clinic will be trained in screening potential participants, questionnaire administration, and data collection. They will also be trained in appropriate informed consent practices. Laboratory study personnel at CDC's Clinical and Environmental Microbiology Branch will also be trained in the handling, preparation, storage, and testing of biologic (stool) specimens.

We do not anticipate inter-observer differences due to the structured and closed-ended format of the questionnaires and the standardization of biologic (stool) specimen collection and testing.

#### **Data Handling and Analysis**

# **Data Collection**

Data from the screening questionnaire and pre-travel questionnaire will be collected on paper and put into REDCap by Dr. Connor's team. Data from the during travel and post-travel questionnaires will be collected electronically (web-based). Red Cap's electronic app (web-based) will be used to collect daily questionnaire data during travel, with an option to have a paper-based form if the participant prefers. Participants will be notified during consent that they should only agree to use web-based data collection during travel if they can reasonably assume that they will have reliable daily internet access; if not, they will be offered paper copies with coded labels. All data collected (either web-based or paper based) will be coded and will be entered and maintained in an electronic database and stored on a secure server by study personnel at The New York Center for Travel and Tropical Medicine clinic.

# Biologic (Stool) Specimen Collection and Testing

Most biologic (stool) specimens will be self-collected by the participant using the DNA Genotek OMNIgene gut kit that will be provided to them at their pre-travel consultation/enrollment visit (each participant will receive 2 kits; one for a pre-travel biologic (stool) specimen and the other for the post-travel biologic [stool] specimen). Each kit includes detailed instructions on collection. All biologic [stool] specimens collected at home will be submitted by mail (postage pre-paid) to the travel clinic. The OMNIgene kits are stable at ambient temperatures for long periods of time and designed for home collection and postal return. Specimens will be mailed from the travel clinic to the CDC's Clinical and Environmental Microbiology Branch in batches. Biologic (stool) specimens will be stored at ambient temperature until DNA extraction.

For those participants able to provide a biologic (stool) sample during their pre-travel clinic consultation/enrollment visit or during a non-study post-travel follow-up sick visit within 10 days of return, study personnel at The New York Center for Travel and Tropical Medicine will aliquot the specimens (see Laboratory Instruments).

All biologic (stool) specimen results will be securely shared through password protected, coded data files. The Clinical and Environmental Microbiology Branch Branch will receive and share only coded information with the co-PIs (see Provision for Protecting Privacy/Confidentiality).

The following analyses will be performed on biologic (stool) specimens collected using the OMNIgene gut kit.

- 1. DNA extraction from single aliquots of stool
- 2. Highly multiplexed PCR assay detecting over 500 different antimicrobial resistance (AMR) genes will be used to test the extracted DNA
- 3. Amplicons produced by the panel will be sequenced on an Illumina MiSeq

Remaining biologic (stool) specimens and extracted DNA will be stored at CDC in the Clinical and Environmental Microbiology Branch indefinitely for potential further use. Stools collected at the clinic and aliquoted for freezing will be stored for potential

further use in analyses that are yet to be determined. Consent for storage of specimens for future research use will be obtained from participants.

#### Provision for Protecting Privacy/Confidentiality

The identity of all study participants will be protected. All questionnaires will be coded using study and group IDs and participants will each be given a unique study ID and group ID. The unique study ID will include a site letter designation of "T", year, and participant number (provided numerically from 1 to 10,000). For example, the unique identifier for the first participant would be: T2017-00001. The group ID will begin with "G" and group number (provided numerically from 1 to 10,000). Those participants who are travel companions and have identical itineraries to other participants in the study and anticipate performing the same activities, (including family and friends), are given the same group number. For example, the group ID for the first participant would be G-00001. If they have a companion traveling with them, that participant would also be G-00001.

The original completed screening questionnaires and any original completed paper daily travel forms will be housed at the clinic in a secure location and destroyed per institutional guidelines.

Biologic (stool) specimens submitted by the participant will be coded. Labels will be provided to the participants for labeling the specimens and will include the participant's unique study ID and group ID. Specimens will be sent to the CDC Clinical and Environmental Microbiology Branch by the Center for Travel and Tropical Medicine for testing and storage.

Labels will also be provided to participants for the paper copies of the during travel questionnaire to ensure confidentiality and to avoid mislabeling.

The database will be password-protected and only study personnel at New York Center for Travel and Tropical Medicine clinic will have access to the password (and thus patient identifiers). No study personnel from CDC will have access to participant identifying information. Identifying information will be stored in a secure, passcode

protected file on a password protected computer and server. This file will be destroyed upon completion of the study.

# <u>Information Management and Analysis Software</u>

Data will be managed securely in REDCap.

SAS v9.4 will be used for analysis.

# Data Entry, Editing and Management, and Data Storage

The New York Center for Travel and Tropical Medicine clinic will be responsible for managing the questionnaire data in REDCap. The data will belong to The New York Center for Travel and Tropical Medicine, will be responsible, in collaboration with partners, for the reporting of findings. Data (questionnaires) done on paper will be stored confidentially at the clinic site and electronic data will be stored confidentially on the REDCap server (see Provision for Protecting Privacy/Confidentiality). The New York Center for Travel and Tropical Medicine clinic will have full access rights and CDC will have access to data (all de-identified) only with the approval of Dr. Connor and his team.

Coded laboratory data in a password-protected database, using the participant's unique ID, will be sent from the laboratory to the New York Center for Travel and Tropical Medicine for input into REDCap.

# **Quality Control and Assurance**

Data quality will be controlled by input of data from screening questionnaires and paper copies of the during travel questionnaires into REDCap by one or two trained personnel at The New York Center for Travel and Tropical Medicine. We will place all data, exactly as received into the database. Data from the web-based questionnaires will be input directly into the REDCap database. Data will not be altered in any way.

Laboratory quality control will be performed by the study laboratorians to ensure that all specimens are tested with appropriate controls as necessary and applicable.

Every 3 months, data entered into REDCap will be checked for completeness and accuracy by the co-PIs (CDC would only access coded data) and/or study personnel; interim data analysis will be performed every 3 months as desired.

#### Bias in Data Collection, Measurement, and Analysis

Double-blinded randomization will control for the introduction of selection bias or observer bias in the study; the participants and the healthcare providers will not know which arm of the study the participant is assigned to. However, our inclusion criteria necessitate the exclusion of travelers with chronic gastrointestinal diseases or travelers on certain medications, possibly creating an exclusion bias. These biases will be addressed in the limitations section of the manuscript. Participants may also introduce recall bias during the pre- and post-travel questionnaires. Reporting bias will be minimized by limiting P&G's involvement with any aspects of the study design, implementation, or analysis.

# **Study Limitations**

As mentioned, a study limitation is the possible incorporation of exclusion bias by excluding travelers with certain chronic medical conditions and those who take certain medications. This will lead to a need to caveat the results of our study to a particular population if the intervention disproves the null hypotheses.

An additional limitation is the inability to collect biologic (stool) samples from participants while abroad in the event that they acquire TD. The collection and sending of biologic (stool) specimens over country borders is complicated and impedes us from collecting real-time potentially infectious specimens to assess the secondary objective — the direct relation between an episode of TD and the acquisition of gut AMR genes.

Participants in the intervention arm of the study may experience side effects of BSS (dark stool and dark discoloration of the mouth) due to oxidization of the bismuth component of the drug. Those in the placebo arm will likely not experience such effects, and the appearance of these effects may cause participants to suspect they were randomized into the intervention arm. Knowledge or suspicion of a participant's own study arm could influence responses to the questionnaire questions.
The results from this study may not be generalizable to all international travelers. This is due to various host factors beyond the study's control and also due to the exclusion of travelers going to regions outside of Asia and Africa. Participants are being recruited from those who are seeking specialized pre-travel medical advice. Not all travelers to the targeted regions seek this care, and travelers who seek pre-travel care may be more likely to comply with safe food/water recommendations. However, by focusing the study on a population of travelers that are visiting places with a high prevalence of TD, the study objectives are likely to be met quickly.

The laboratory assays also have limitations. The multiplex PCR assay detecting AMR genes will not provide any information regarding the organism of origin for the genes detected, including whether or not two or more genes originated from the same organism or if multiple organisms harbor the same resistance gene. This assay is only capable of detecting genes for which primers are included in the assay. However, the assay currently includes more than 500 targets and can be expanded to include additional targets of interest to study stakeholders. Also, many of the primers on this panel will readily amplify closely related gene variants even if a specific primer pair is not present, e.g. a *tetX* primer pair may amplify a *tetA* gene. Finally, the presence of a specific gene product does not guarantee the gene itself is expressed as functional antimicrobial resistance.

An additional limitation is that culture cannot be obtained from most biologic (stool) samples, making it difficult to answer future questions that involve assigning AMRs to particular organisms, unless there are further advances in sequencing/bioinformatic technology. Without a pre-screening step like the highly multiplexed PCR assay suggested, the scope of the study will have to be significantly limited to a few AMR gene groups because the real time isolation and testing of samples as they are collected is labor intensive and cannot include the breadth of targets possible with molecular testing.

Response to New or Unexpected Findings and Changes in the Study Environment

If a new or unexpected finding is identified, the co-PIs and collaborating partners will be alerted immediately. Depending on the scope and potential morbidity associated with this finding, appropriate action will be taken.

Additionally, an incident report will be filed as required by the reviewing IRB if there is an unexpected violation of study procedures or expectations or if unanticipated problems or adverse events are identified.

If deemed necessary by the IRB, we would consider using a Study Data Safety Monitoring Board to analyze the data and stop the study early in the event there are serious adverse outcomes that are significantly higher in the placebo or intervention arm. However, due to the relative safety of BSS, we do not anticipate this will be necessary.

Due to the number of participants that will need to be enrolled in this study to achieve adequate power, there is the possibility that this study may extend beyond the current study timeline. Although we do not anticipate difficulty enrolling participants, we want be prepared for any unanticipated issues with enrollment. In the event that 488 participants are not enrolled at two years, an interim analysis will be performed and additional funding will be requested to continue the project until adequate power is achieved.

#### <u>Identifying, Managing, and Reporting Adverse Events</u>

Adverse events in this study may include, but are not limited to, the following:

- 1. Medication side effects, such as constipation, tinnitus, or dizziness
- Medication adverse events, such as neurologic findings from salicylate toxicity (confusion, slurred speech, drowsiness, muscle weakness, headache, mental depression) or severe stomach pain, increased sweating, or increased thirst

All participants will be asked about adverse events on each of the study questionnaires, including the daily questionnaire while traveling. If the participant experiences an

adverse event while abroad, they are to stop the study medication and contact the study personnel to report the symptoms and obtain advice.

### Notifying Participants of their Individual Results

Participants will not be notified of their study results, since the results will not impact their healthcare.

## **Disseminating Information to the Public**

The results from this study will be published in a peer-reviewed journal, however, the initial release may be in the form of an abstract for a scientific meeting.

Preliminary study findings will be shared with P&G after the data analysis phase is complete.

# **Budget Estimates**

Table 4. CLINIC events with estimated costs (primary objective)

NOTE: Table 4 costs are for 500 participants

| | Pre-travel consultation/ enrollment visit (baseline) | During travel | Post-travel | TOTAL |
|---|---|---|---|---|
| Recruitment materials | \$200 | N/A | N/A | \$200 |
| Printing costs (screening | \$50 | \$150 | N/A <sup>a</sup> | \$200 |
| questionnaire, daily travel | | | | |
| logs, labels) | | | | |
| Participant compensation | \$100 per participant | up to \$100 per<br>participant<br>(\$5 per entry) | \$100 per<br>participant | \$150,000 |
| Advertising | \$1,500 | N/A | N/A | \$1,500 |
| IRB Costs | \$3,000 | N/A | N/A | \$3,000 |
| Prepaid envelopes for | N/A | \$1,000 (\$2.00 stamp) | N/A | \$1,000 |
| during-travel questionnaires | | | | |
| Shipment of study medications from CDC to | \$10,000 | N/A | N/A | \$10,000 |
| clinic | | | | |
| Administrative Personnel Costs: Physician | \$110,000 | N/A | N/A | \$110,000 |
| PI (5%) plus study | | | | |
| coordinator (40%) | | | | |
| Recruitment/enrollment, | | | | |
| documentation and | | | | |
| completion of study forms | | | | |
| and participant and data | | | | |
| follow up | | | | |
| Travel (conferences) | N/A | N/A | \$20,000 | \$20,000 |

| TOTAL | \$295,900 |
|-------|-----------|

<sup>&</sup>lt;sup>a</sup>Not applicable

Table 5. LABORATORY events with estimated costs

| | Stages | | | |
|---|---|---|---|---|
| | Pre-travel | During travel | Post-travel | TOTAL |
| | consultation/enrollment | | | |
| | visit (baseline) | | | |
| Supplies for stool sample | \$25 | N/A | \$25 | \$25,000 |
| (OMNIgene gut kit) | | | | |
| (n=1,000 stools or 500 participants) | | | | |
| Shipping stool sample to the clinic | \$10 per sample | N/A | \$10 per | \$10,000 |
| (n=1,000 stools or 500 participants) | | | sample | |
| Shipping stool samples to CDC lab | \$15 per sample | N/A | \$15 per | \$15,000 |
| from clinic | | | sample | |
| (n=1,000 stools or 500 participants) | | | | |
| Diagnostic testing of stool | | | | |
| (n=500 stools or 250 participants) | | | | |
| DNA extraction | \$15 | N/A | \$15 | \$7,500 |
| PCR (AMR gene assay) | \$35 | N/A | \$35 | \$17,500 |
| Amplicon sequencing | \$25 | N/A | \$25 | \$12,500 |
| Laboratorian (ORISE) | \$28,000 | N/A | N/A | \$28,000 |
| Bioinformatics (ORISE) | \$66,000 | N/A | N/A | \$66,000 |
| TOTAL | | | | \$181,500 |

Table 6. Cumulative costs of both CLINIC and LABORATORY events from Table 4 and Table 5

| Cumulative totals | Total |
|-------------------|-----------|
| Clinic Events | \$295,900 |
| Laboratory Events | \$181,500 |
| | \$477,400 |

### References

- 1. Connor B. Travelers' diarrhea. In Yellow Book (pp. 60-64). New York, NY: Oxford University Press; 2016.
- 2. Brum J, Gibb R, Ramsey D, Balan G, Yacyshyn B. Meta-analyses assessment of the clinical efficacy of bismuth subsalicylate for prevention and treatment of infectious diarrhea. [not yet published]
- 3. DuPont HL, Ericsson CD, Johnson PC, de la Calabra. Use of bismuth subsalicylate for the prevention of travelers' diarrhea. *Rev Infect Dis*, 1990; Suppl 1:S67–67.
- 4. DuPont HL, Ericsson CD, Johnson PC, Bitsura JM, DuPont MW, de la Cabada FJ. Prevention of travelers' diarrhea by tablet formulation of bismuth subsalicylate. *JAMA*, 1987; 257(10):1347–1350.
- 5. Steffen R, DuPont HL, Huesser R, Helminger A, Witassek F, Manhart MD, Schär M. Prevention of travelers' diarrhea by the tablet form of bismuth subsalicylate. *Antimicrob Agents Chemother*, 1986; 29:625–629.
- 6. Graham DY, Estes MK, Gentry LO. Double-blind comparison of bismuth subsalicylate and placebo in the prevention and treatment of enterotoxigenic *Escherichia coli*-induced diarrhea in volunteers.

  \*\*Gastroenterology\*, 1983; 85(5):1017–1022.
- 7. Reynolds PT, Abalos KC, Hopp J, Williams ME. Bismuth toxicity: a rare cause of neurologic dysfunction. *Int J Clin Med*, 2012; 3:46–48.
- 8. Gordon MF, Abrams RI, Rubin DB, Barr WB, Correa DD. Bismuth subsalicylate toxicity as a cause of prolonged encephalopathy with myoclonus. *Mov Disord*, 1995; 10(2):220–222.
- 9. Pitz AM, Park GW, Lee D, Boissy YL, Vinjé J. Antimicrobial activity of bismuth subsalicylate on *Clostridium difficile*, *Escherichia coli* O157:H7, norovirus, and other common enteric pathogens. *Gut Microbes*, 2015; 6(2):93–100.
- 10. Manhart MD. In vitro antimicrobial activity of bismuth subsalicylate and other bismuth salts. *Rev Infect Dis*, 1990; 21 Suppl 1, S11–15.
- 11. Sox TE, Olson CA. Binding and killing of bacteria by bismuth subsalicylate. *Antimicrob Agents Chemother*, 1989; 33(12):2075–2082.
- 12. Ericsson CD, Evans DG, DuPont HL, Evans DJ Jr, Pickering LK. Bismuth subsalicylate inhibits activity of crude toxins of *Escherichia coli* and *Vibrio cholerae*. *J Infect Dis*, 1977; 136(5):693–696.
- Centers for Disease Control and Prevention. Antibiotic Resistance Threats in the United States, 2013.
   Available at: <a href="https://www.cdc.gov/drugresistance/pdf/ar-threats-2013-508.pdf">https://www.cdc.gov/drugresistance/pdf/ar-threats-2013-508.pdf</a> Accessed 22 March 2017.
- 14. Hassing RJ, Alsma J, Arcilla MS, van Genderen PJ, Stricker BH, Verbon A. International travel and acquisition of multidrug-resistant Enterobacteriaceae: a systematic review. *Euro Surveill*, 2015; 20(47).

- 15. Ruppé E, Armand-Lefevre L, Estellat C, Consigny PH, El Mniai A, Boussadia Y, Goujon C, Ralaimazava P, Campa P, Girard PM, Wyplosz B, Vittecog D, Bouchard O, Le Loup G, Pialoux G, Perrier M, Wieder I, Moussa N, Esposito-Farèse M, Hoffmann I, Coignard B, Lucet JC, Andremont A, Matheron S. High rate of acquisition but short duration of carriage of multidrug-resistant Enterobacteriacae after travel to the tropics. *Clin Infect Dis*, 2015; 61(4):593–600.
- 16. Angue M, Allou N, Belmonte O, Lefort Y, Lugagne N, Vandroux D, Montravers P, Allyn J. Risk factors for colonization with multidrug-resistant bacteria among patients admitted to the intensive care unit after returning from abroad. *J Travel Med*, 2015; 22(5): 300–305.
- 17. Epelboin L, Robert J, Tsyrina-Kouyoumdjian E, Laouira S, Meyssonnier V, caumes E. High rate of multidrug-resistant gram-negative bacilli carriage and infection in hospitalized returning travelers: a cross-sectional cohort study. *J Travel Med*, 2015; 22(5): 292–299.
- 18. Arcilla MS, van Hattem JM, Haverkate MR, et al. Import and spread of extended-spectrum β-lactamase-producing Enterobacteriaceae by international travellers (COMBAT study): a prospective, multicentre cohort study. *Lancet Infect Dis*, 2017; 17(1): 78-85.
- 19. Kantele A. A call to restrict prescribing antibiotics for travellers' diarrhea Travel medicine practitioners can play an active role in preventing the spread of antimicrobial resistance. *Trav Med Infect Dis*, 2015; 13(3): 213.
- 20. Bowen A, Agboatwalla M, Pitz AM, Brum J, Plikaytis B. Bismuth subsalicylate reduces antimicrobial medication use among adult diarrhea outpatients in Pakistan: a randomized, placebo-controlled, triplemasked clinical trial. ASTMH 65th Annual Meeting. Atlanta, Georgia, 2016.
- 21. World Tourism Organization. UNWTO tourism highlights: 2014 edition. Available at: <a href="http://mkt.unwto.org/publication/unwto-tourism-highlights-2014-edition">http://mkt.unwto.org/publication/unwto-tourism-highlights-2014-edition</a>. Accessed 9 March 2017.
- 22. World Health Organization. Antimicrobial Resistance Global Report on Surveillance. 2014. Available at: <a href="http://apps.who.int/iris/bitstream/10665/112642/1/9789241564748\_eng.pdf">http://apps.who.int/iris/bitstream/10665/112642/1/9789241564748\_eng.pdf</a>. Accessed 15 March 2017.
- 23. Hassing RJ, Alsma J, Arcilla MS, van Genderen PJ, Stricker BH, Verbon A. International travel and acquisition of multidrug-resistant Enterobacteriaceae: a systematic review. *Euro Surv*, 2015; 20(47).
- 24. Von Wintersdorff CJH, Penders J, Stobberingh EE, et al. High rates of antimicrobial drug resistance gene acquisition after international travel, the Netherlands. *Emerg Infect Dis*, 2014; 20(4):649–657.
- 25. Connor BA. Sequelae of traveler's diarrhea: focus on post-infectious irritable bowel syndrome. *Clin Infect Dis*, 2005; 41(8): S577–586.
- 26. Bierer DW, Bismuth subsalicylate: history, chemistry, and safety. Rev Infect Dis, 1990; 12(1):3-8.

| 27. | 27. Ericsson CD, Feldman S, Pickering LK, Cleary TG. Influence of subsalicylate bismuth on absorption of |
|---|---|
| | doxycycline. JAMA, 1982; 247(16):2266–2267. |

## APPENDIX A: Screening Questionnaire



### **Screening Questionnaire**

Script [read to all travelers]: Hello, my name is [name] and I am a [role in the clinic] at The New York Center for Travel and Tropical Medicine. We are conducting a study of international travelers to see if bismuth subsalicylate (or BSS) can help to prevent travelers' diarrhea. Participation in this questionnaire to see if you are eligible is voluntary, and it will only take a moment of your time. We will be collecting your email address, so in the event that you are eligible to participate, we can send you the study questionnaires and reminder emails; your email will only be used for study purposes. Are you interested in seeing if you are eligible to participate?

| [If "yes", please complete the fo | ollowing with the travel | er]: | |
|---|---|---|---|
| Participant's Initials | | Date | |
| Age | | | |
| ☐ Participant Email (REQUIRED): | | | |
| ☐ Participant Phone #1 (OPTIONAL | | rticipant Phon | e #2 (OPTIONAL): |
| <ol> <li>Are you ≥ 18 years of age and </li> </ol> | <70 years of age? | | |
| ☐ Yes* | □ No | | ☐ Don't know |
| 2. Are you traveling to either Sou | | al Asia, North | |
| ☐ Yes* | □ No | | ☐ Don't know |
| s. Are you spending at least 7 day | ys and no more than 21 da | ays in these re | egions? |
| ☐ Yes* | □ No | | ☐ Don't know |
| . Are you leaving for your trip in | at least 7 days? | | |
| ☐ Yes* | □ No | | ☐ Don't know |
| i. Are you now pregnant or nursi | ng or do you plan to get p | regnant befo | re the end of your trip? |
| □ Yes | □ No* | | ☐ Don't know |

| Do you have kno | own or suspected | ancigy to bisinatil, salicyla | te, or aspirin: |
|---|---|---|---|
| □ Y | es | □ No* | ☐ Don't know |
| - | • | allergy to microcrystal cellusaccharin, or talc? | ulose, calcium carbonate, artificial coloring, |
| □ Y | es | □ No* | ☐ Don't know |
| Do you have kid | ney disease, diabo | etes, gout, or a clotting disc | order? |
| □ Y | es | □ No* | ☐ Don't know |
| - | <ul><li>an antibiotic in th</li><li>Doxycycline or</li></ul> | ne past 30 days? For exampler minocycline | le: |
| | | oxazole (e.g., Bactrim, Septr | a) |
| | <ul> <li>Penicillins (e.g</li> </ul> | g., amoxicillin, Augmentin) | |
| | | ns (e.g., Keflex) | |
| | • | nes (e.g., ciprofloxacin) | |
| | <ul> <li>N/aavalidaa/a</li> </ul> | | 1 (1 |
| | • Macrolides (e. | g., azithromycin [Zithromax | g, erythromycin) |
| □ Y | | g., azitnromycin (zitnromax | □ Don't know |
| □ Y | es | □ No* | |
| □ Y | es<br>of the following I | □ No* medications or therapies? | |
| □ Y Do you take any | es of the following i Chronic oral of steroids | □ No* medications or therapies? | ☐ Don't know g., hydrocortisone or prednisone); not inhaled |
| □ Y<br>Do you take any | of the following age. Alkylating age. Antimetabolite | □ No* medications or therapies? r intravenous IV steroids (e. nts (e.g., cyclophosphamide | Don't know g., hydrocortisone or prednisone); not inhaled e [Cytoxan]) an], 6-mercaptopurine [Purinethol]) |
| □ Y Do you take any | of the following of the | □ No* medications or therapies? r intravenous IV steroids (e. nts (e.g., cyclophosphamide es (e.g., azathioprine [Imura eutic agents (e.g., including is factor (TNF) blockers (e.g. | Don't know g., hydrocortisone or prednisone); not inhaled e [Cytoxan]) an], 6-mercaptopurine [Purinethol]) |
| □ Y | es of the following of | □ No* medications or therapies? r intravenous IV steroids (e. nts (e.g., cyclophosphamide es (e.g., azathioprine [Imura eutic agents (e.g., including is factor (TNF) blockers (e.g.) pegol [Entyvio], golimumab | Don't know g., hydrocortisone or prednisone); not inhaled e [Cytoxan]) an], 6-mercaptopurine [Purinethol]) methotrexate [Trexall]) ., etanercept [Enbrel], adalimumab [Humira], |
| □ Y | es of the following in | □ No* medications or therapies? r intravenous IV steroids (e. nts (e.g., cyclophosphamide es (e.g., azathioprine [Imura eutic agents (e.g., including is factor (TNF) blockers (e.g.) pegol [Entyvio], golimumab | Don't know g., hydrocortisone or prednisone); not inhaled e [Cytoxan]) an], 6-mercaptopurine [Purinethol]) methotrexate [Trexall]) , etanercept [Enbrel], adalimumab [Humira], [Simponi], and infliximab [Remicade]) ituxan] or alemtuzumab [Lemtrada]) |
| □ Y | es of the following of | □ No* medications or therapies? r intravenous IV steroids (e. nts (e.g., cyclophosphamide es (e.g., azathioprine [Imura eutic agents (e.g., including is factor (TNF) blockers (e.g. pegol [Entyvio], golimumab ntibodies (e.g., rituximab [R lumalog, NPH, Lantus, Lever e.g., divalproex, Depakote, | Don't know g., hydrocortisone or prednisone); not inhaled e [Cytoxan]) an], 6-mercaptopurine [Purinethol]) methotrexate [Trexall]) and etanercept [Enbrel], adalimumab [Humira], [Simponi], and infliximab [Remicade]) ituxan] or alemtuzumab [Lemtrada]) mir) Depacon) |
| □ Y | es of the following in | □ No* medications or therapies? r intravenous IV steroids (e. nts (e.g., cyclophosphamide es (e.g., azathioprine [Imura eutic agents (e.g., including is factor (TNF) blockers (e.g. pegol [Entyvio], golimumab ntibodies (e.g., rituximab [R lumalog, NPH, Lantus, Lever e.g., divalproex, Depakote, s (e.g., lisinopril [Zestril], ena zepril [Lotensin]) | Don't know g., hydrocortisone or prednisone); not inhaled e [Cytoxan]) an], 6-mercaptopurine [Purinethol]) methotrexate [Trexall]) ., etanercept [Enbrel], adalimumab [Humira], [Simponi], and infliximab [Remicade]) ituxan] or alemtuzumab [Lemtrada]) mir) Depacon) alapril [Vasotec], captopril [Capoten], ramipril |
| □ Y | es of the following of | □ No* medications or therapies? r intravenous IV steroids (e. nts (e.g., cyclophosphamide es (e.g., azathioprine [Imura eutic agents (e.g., including is factor (TNF) blockers (e.g. pegol [Entyvio], golimumab ntibodies (e.g., rituximab [R lumalog, NPH, Lantus, Lever e.g., divalproex, Depakote, s (e.g., lisinopril [Zestril], ena zepril [Lotensin]) | Don't know g., hydrocortisone or prednisone); not inhaled e [Cytoxan]) an], 6-mercaptopurine [Purinethol]) methotrexate [Trexall]) and infliximab [Remicade]) ituxan] or alemtuzumab [Lemtrada]) mir) Depacon) alapril [Vasotec], captopril [Capoten], ramipril l, aspirin, clopidogrel [Plavix], argatroban |

# 11. Do you have any of the following chronic stomach or intestinal illnesses?

- Irritable bowel syndrome (IBS)
- Inflammatory bowel disease (including ulcerative colitis and Crohn's disease)
- Celiac disease; any form of chronic diarrhea or chronic abdominal pain;
- Pancreatic insufficiency
- Gallbladder disease
- Malabsorption syndromes
- Gastrointestinal malignancy/cancer currently receiving chemo; radio, or immunotherapy
- Chronic diarrhea from another cause

| | ☐ Yes | □ No* | | ☐ Don't know |
|---|---|---|---|---|
| 12. Do | you have any illne<br>Missing or non-fu | sses that you have been told I | owers your body | y's ability to fight infection? |
| • | Insulin-dependent | | edications (e.g. r | netformin, glyburide) |
| • | deficiency) | iciency syndrome (e.g. comple | | |
| | immunocomprom | | | ap,, o. a.,, oe. |
| | ☐ Yes | □ No* | | ☐ Don't know |
| 13. Ha | ave you ever receive | ed a solid organ transplant? | | |
| | ☐ Yes | □ No* | | ☐ Don't know |
| | cu currently have dia | □ No* | ' to all subsequei | □ Don't know<br>nt to be eligible for enrollment. |
| □ Eli | gible per Appx A | ☐ Not Eligible per Appx A | Comments: | |
| By signing below, I confirm that I conducted the verbal screening and have reviewed the answers before proceeding with additional study activities: | | | | |
| Nam | e of Interviewer | | Signature | |
| Date | | | | |
| If elig | ible, collect the fol | lowing: | | |
| State o | pant First Name:<br>of Residence:<br>ence Zip Code: | County of Residence | | Name: |
| Genei | ration of Study ID a | and Group ID: | | |

### **UNIQUE STUDY ID:**

The unique study ID will include a site letter designation of "T", year, and participant number (provided numerically from 1 to 10,000).

\*For example, the unique identifier for the first participant would be: T2017-00001.

### **GROUP ID:**

The group ID will begin with "G" and a group number (provided numerically from 1 to 10,000). Those participants who are travel companions and have identical itineraries to other participants in the study

and anticipate performing the same activities, (including family and friends), are given the same number.

\*For example, the group ID for the first participant would be G-00001. Their mother, traveling with them, would also be G-00001.

| 6. 1 15.41 |
|-------------------|
| Study ID Number |
| Study ID Italiaci |
| 1 |

# APPENDIX B: Country Listing for Inclusion

### **South East Asia**

| Cambodia |
|--------------------------------------------|
| Laos |
| West Malaysia (excluding Malaysian Borneo) |
| Myanmar (Burma) |
| Thailand |
| Vietnam |

## **South Central Asia**

| Afghanistan |
|-------------|
| Bangladesh |
| Bhutan |
| India |
| Maldives |
| Nepal |
| Pakistan |
| Sri Lanka |

## **North Africa**

| Algeria | |
|---------|---|
| Egypt | |
| Libya | |
| Morocco | |
| Sudan | _ |
| Tunisia | |

# Sub-Saharan Africa (Does NOT include the country of SOUTH AFRICA)

| Angola | Congo | Guinea-Bissou | Mozambique | Sierra Leone |
|---|---|---|---|---|
| Benin | Democratic Republic | Kenya | Namibia | Somalia |
| | of the Congo | | | |
| Botswana | Côte d' Ivoire | Lesotho | Niger | South Sudan |
| Burkina Faso | Djibouti | Liberia | Nigeria | Swaziland |
| Burundi | Equatorial Guinea | Madagascar | Reunion | United Republic of |
| | | | | Tanzania |
| Cameroon | Eritrea | Malawi | Rwanda | The Gambia |
| Cabo (Cape) Verde | Ethiopia | Mali | Saint Helena | Togo |
| Central African | Gabon | Mauritania | São Tomé and | Uganda |
| Republic | | | Príncipe | |
| Chad | Ghana | Mauritius | Senegal | Zambia |
| Comoros | Guinea | Mayotte | Seychelles | Zimbabwe |



# **Pre-travel Questionnaire**

| | PARTICIPANT UNIQUE ID: |
|---|---|
| | GROUP ID: |
| [Please rev | view the screening questionnaire with the participant.] |
| = | be been any changes to the screening questionnaire making the participant ineligible to participate? |
| | Yes |
| b. | No |
| If yes, plea | se describe: |
| Demograp | hics |
| Age (in yea | nrs): |
| Sex (M/F): | |
| Race: | |
| _ | White or Caucasian |
| | Black or African American |
| | American Indian or Alaskan native |
| | Asian or Pacific Islander |
| | Other (please specify) |
| | Don't know |
| g. | I would rather not answer |
| Ethnicity: | |
| a. | Hispanic |
| b. | Non-Hispanic |
| Medical Hi | story |
| - | a have any medical conditions or illnesses? |
| a. | Yes |
| | No |
| _ | Don't know |
| d. | I would rather not answer |
| If yes t | o question 1, please list them all. |

| 3. Do you | have recurrent or persistent tinnitus (ringing in the ears)? |
|-----------|--------------------------------------------------------------|
| a. | Yes |
| b. | No |
| C. | Don't know |
| d. | I would rather not answer |

- 4. Do you take any medications on a regular basis?
  - a. Yes
  - b. No
  - c. Don't know
  - d. I would rather not answer

#### If Yes to guestion 3, please list them all:

| 1. | 4. |
|----|----|
| 2. | 5. |
| 3. | 6. |

- 5. Have you taken any oral or intravenous (IV) antibiotics in the past 90 days for any reason (e.g., azithromycin [Zithro-max], ciprofloxacin [Cipro], rifaximin [Xifaxan], doxycycline or minocycline, metronidazole [Flagyl], cotrimoxazole [Bactrim or Septra], penicillins [e.g., amoxicillin or Augmentin], or cephalosporins [e.g., Keflex])?
  - a. Yes
  - b. No
  - c. Don't know
  - d. I would rather not answer

#### If yes to question 4, please give the antibiotic name, start date, duration, and illness taken for:

| No. | Antibiotic Name | Start Date<br>(MM/DD/YYYY) | Duration<br>(Days) | Illness taken for |
|---|---|---|---|---|
| 1 | | | | |
| 2 | | | | |
| 3 | | | | |
| 4 | | | | |
| 5 | | | | |
| 6 | | | | |

### 6. In the past 30 days, have you taken a probiotic? -

Probiotics are live microorganisms (such as certain types of bacteria) that may benefit the health of the person consuming them. Yogurts and other fermented dairy products are probiotics. Probiotics can also take the form of capsules, pills, or powders. Probiotics also include any foods or drinks labeled as containing "live and active cultures" or "probiotics."

a. Yes

- b. No
- c. Don't know
- d. I would rather not answer

### **Travel History**

- 7. Have you traveled internationally in the past 90 days?
  - a. Yes
  - b. No
  - c. Don't know
  - d. I would rather not answer

If yes to question 6, which countries did you travel to and what were your dates of travel? If the exact dates of travel are unknown, please list the month and year only.

| dates of travel are unknown, please list the month and yea | |
|---|---|
| Country name | Dates of travel<br>(MM/DD/YY to<br>MM/DD/YY) |
| 1. | // to//_ |
| 2. | // to//_ |
| 3. | // to// |
| 4. | // to//_ |
| 5. | // to// |
| 6. | // to//_ |

8. Where are you planning to travel? Please specify each country name, the specific locations you plan to visit, and the number of days you plan to spend in each country.

| Country name | Specific location(s) to be visited (e.g., city/town, attraction) | Number of days in this country |
|---|---|---|
| 1. | | |
| 2. | | |
| 3. | | |

| 4. |
|----|
| 5. |
| 6. |

#### 9. What is the total duration of your trip (in days)?

\_\_\_\_\_

### 10. What is your main reason for travel (circle only one)?

- a. Education or research (includes medical or veterinary-type education)
- b. Adoption
- c. Business
- d. Leisure/tourism
- e. Immigrant traveling back to visit friends or relatives
- f. Providing medical care as a health professional (including paid or unpaid/volunteer)
- g. Receiving medical care (as a patient)
- h. Non-medical service or volunteer work
- i. Missionary work
- j. Military service
- k. Attending large gathering or event (e.g., large sporting event, large conference, Hajj)
- 1. Adventuring (extreme mountaineering, water sports, outdoor activities, etc.)
- m. Other:

\_\_\_\_\_

n. I would rather not answer

#### 11. What are the secondary reasons for travel (circle all that apply)?

- a. Education or research (includes medical or veterinary-type education)
- b. Adoption
- c. Business
- d. Leisure/tourism
- e. Returning to region of origin of self or family to visit friends and relatives
- f. Providing medical care as a health professional (including paid or unpaid/volunteer)
- g. Receiving medical care (as a patient)
- h. Non-medical service or volunteer work
- i. Missionary work
- j. Military service
- k. Attending large gathering or event (e.g., large sporting event, large conference, Hajj)
- I. Adventuring (extreme mountaineering, water sports, outdoor activities, etc.)
- m. Other:

\_\_\_\_\_

n. I would rather not answer

Thank you very much for your time.

# APPENDIX D: During-travel Questionnaire

# **During Travel Questionnaire**

| PARTICIPANT UNIQUE ID: |
|------------------------|
| GROUP ID: |
| GROUP ID: |

| | Day 1 | Day 2 | Day 3 | Day 4 | Day 5 |
|---|---|---|---|---|---|
| Please write the calendar date that corresponds to each day of your trip. | | | | | |
| Day 1 is your first day of arrival in the country. | | | | | |
| Number of tablets taken in the morning (maximum 4) | | | | | |
| Number of tablets taken in the afternoon/evening (maximum 4) | | | | | |
| Symptoms in the prior 24 hours (check off all that apply) | | | | | |
| Fever | | | | | |
| Nausea | | | | | |
| Vomiting | | | | | |
| Loose stools (less than three in a 24 hour period) | | | | | |
| Diarrhea (three or more loose stools in 24 hours) | | | | | |
| Bloody diarrhea | | | | | |
| Constipation | | | | | |
| Dark or black stool | | | | | |
| Dark or black tongue | | | | | |
| Abdominal pain | | | | | |
| Abdominal cramps | | | | | |
| Urgency to relieve oneself (in reference to stool) | | | | | |
| Bloating | | | | | |
| Flatulence/gas | | | | | |
| Congestion/runny nose | | | | | |
| Sore throat | | | | | |
| Cough | | | | | |
| Rash | | | | | |
| Headache | | | | | |
| Dizziness | | | | | |
| Ringing in your ears | | | | | |
| Muscle pain/soreness | | | | | |
| loint nain/swelling/redness | П | П | П | | П |

| Drowsiness (severe) | | | | | |
|---|---|---|---|---|---|
| Confusion | | | | | |
| Depression | | | | | |
| Other (list/describe): | | | | | |
| Medical care | | | | | |
| Did you seek medical care for one or more of these symptoms? | Y N D | Y N D | Y N D | Y N D | Y N D |
| (Yes/No/Don't Know) | | | | | |
| → If yes, where? (check the corresponding box(es)) | | | | | |
| A doctor's office | | | | | |
| Urgent care clinic (outpatient) | | | | | |
| Emergency room | | | | | |
| Hospital outpatient clinic setting | | | | | |
| Hospital inpatient ward – hospitalized | | | | | |
| Other (specify) | | | | | |
| → Was your diagnosis travelers' diarrhea? | Y N D | Y N D | Y N D | Y N D | Y N D |
| (Yes/No/Don't Know) | | | | | |
| Have you started any medications in the past 24 hours? | Y N D | Y N D | Y N D | Y N D | Y N D |
| (Yes/No/Don't Know) | | | | | |
| → If yes, what medication(s)? | | | | | |
| → Please circle those that were provided for you at | | | | | |
| your pre-travel consultation with the study clinic. | | | | | |
| What city(ies) and country(ies) have you been in during the past 24 hours? | | | | | |
| Please write answers to all questions in the corresponding box. | | | | | |
| Have you eaten any of the following in the past 24 hours? | | | | | |
| (Yes/No/Don't Know) | V N D | V N D | V N D | V N D | V N D |
| → Fermented or pickled foods (e.g., bean paste, fish | Y N D | Y N D | Y N D | Y N D | Y N D |
| kimchi, etc.) | V N D | V N D | V N D | V N D | V N D |
| → Yogurt | YND | YND | YND | YND | YND |
| Did you have any diarrhea between completing the pre-travel | Y N D | | | | |
| questionnaire and arriving in the country? (Yes/No/Don't Know) | | | | | |
| Comments: | | | | | |

| PARTICIPANT UNIQUE ID: |
|------------------------|
| GROUP ID: |

| | Day 6 | Day 7 | Day 8 | Day 9 | Day 10 |
|---|---|---|---|---|---|
| Please write the calendar date that corresponds to each day of your trip. Day 1 is your first day of arrival in the country. | | | | | |
| Number of tablets taken in the morning (maximum 4) | | | | | |
| Number of tablets taken in the afternoon/evening (maximum 4) | | | | | |
| Symptoms in the prior 24 hours (check off all that apply) | | | | | |
| Fever | | | | | |
| Nausea | | | | | |
| Vomiting | | | | | |
| Loose stools (less than three in a 24 hour period) | | | | | |
| Diarrhea (three or more loose stools in 24 hours) | | | | | |
| Bloody diarrhea | | | | | |
| Constipation | | | | | |
| Dark or black stool | | | | | |
| Dark or black tongue | | | | | |
| Abdominal pain | | | | | |
| Abdominal cramps | | | | | |
| Urgency to relieve oneself (in reference to stool) | | | | | |
| Bloating | | | | | |
| Flatulence/gas | | | | | |
| Congestion/runny nose | | | | | |
| Sore throat | | | | | |
| Cough | | | | | |
| Rash | | | | | |
| Headache | | | | | |
| Dizziness | | | | | |
| Ringing in your ears | | | | | |
| Muscle pain/soreness | | | | | |
| Joint pain/swelling/redness | | | | | |
| Drowsiness (severe) | | | | | |
| Confusion | | | | | |
| Depression | | | | | |

| Other (list/describe): | | | | | |
|---|---|---|---|---|---|
| other (had describe). | _ | _ | | | |
| Medical care | | | | | |
| Did you seek medical care for one or more of these symptoms? | Y N D | Y N D | Y N D | Y N D | Y N D |
| (Yes/No/Don't Know) | | | | | |
| → If yes, where? (check the corresponding box(es)) | | | | | |
| A doctor's office | | | | | |
| Urgent care clinic (outpatient) | | | | | |
| Emergency room | | | | | |
| Hospital outpatient clinic setting | | | | | |
| Hospital inpatient ward – hospitalized | | | | | |
| Other (specify) | | | | | |
| → Was your diagnosis travelers' diarrhea? | Y N D | Y N D | Y N D | Y N D | Y N D |
| (Yes/No/Don't Know) | | | | | |
| Have you started any medications in the past 24 hours? | Y N D | Y N D | Y N D | YND | Y N D |
| (Yes/No/Don't Know) | | | | | |
| → If yes, what medication(s)? | | | | | |
| → Please circle those that were provided for you at | | | | | |
| your pre-travel consultation with the study clinic. | | | | | |
| What city(ies) and country(ies) have you been in during the past 24 hours? | | | | | |
| Please write answers to all questions in the corresponding box. | | | | | |
| Trease write union to an question in the corresponding now | | | | | |
| Have you eaten any of the following in the past 24 hours? | | | | | |
| (Yes/No/Don't Know) | | | | | |
| → Fermented or pickled foods (e.g., bean paste, fish | Y N D | Y N D | Y N D | Y N D | Y N D |
| kimchi, etc.) | | | | | |
| → Yogurt | Y N D | Y N D | Y N D | Y N D | Y N D |
| Comments: | | | | | |
| Comments. | | | | | |

| PARTICIPANT UNIQUE ID: |
|------------------------|
| GROUP ID: |

| | Day 11 | Day 12 | Day 13 | Day 14 | Day 15 |
|---|---|---|---|---|---|
| Please write the calendar date that corresponds to each day of your trip. Day 1 is your first day of arrival in the country. | | | | | |
| Number of tablets taken in the morning (maximum 4) | | | | | |
| Number of tablets taken in the afternoon/evening (maximum 4) | | | | | |
| Symptoms in the prior 24 hours (check off all that apply) | | | | | |
| Fever | | | | | |
| Nausea | | | | | |
| Vomiting | | | | | |
| Loose stools (less than three in a 24 hour period) | | | | | |
| Diarrhea (three or more loose stools in 24 hours) | | | | | |
| Bloody diarrhea | | | | | |
| Constipation | | | | | |
| Dark or black stool | | | | | |
| Dark or black tongue | | | | | |
| Abdominal pain | | | | | |
| Abdominal cramps | | | | | |
| Urgency to relieve oneself (in reference to stool) | | | | | |
| Bloating | | | | | |
| Flatulence/gas | | | | | |
| Congestion/runny nose | | | | | |
| Sore throat | | | | | |
| Cough | | | | | |
| Rash | | | | | |
| Headache | | | | | |
| Dizziness | | | | | |
| Ringing in your ears | | | | | |
| Muscle pain/soreness | | | | | |
| Joint pain/swelling/redness | | | | | |
| Drowsiness (severe) | | | | | |
| Confusion | | | | | |
| Denression | | | | | |

| Other (list/describe): | | | | | |
|---|---|---|---|---|---|
| other (had describe). | _ | _ | | | |
| Medical care | | | | | |
| Did you seek medical care for one or more of these symptoms? | Y N D | Y N D | Y N D | Y N D | Y N D |
| (Yes/No/Don't Know) | | | | | |
| → If yes, where? (check the corresponding box(es)) | | | | | |
| A doctor's office | | | | | |
| Urgent care clinic (outpatient) | | | | | |
| Emergency room | | | | | |
| Hospital outpatient clinic setting | | | | | |
| Hospital inpatient ward – hospitalized | | | | | |
| Other (specify) | | | | | |
| → Was your diagnosis travelers' diarrhea? | Y N D | Y N D | Y N D | Y N D | Y N D |
| (Yes/No/Don't Know) | | | | | |
| Have you started any medications in the past 24 hours? | Y N D | Y N D | Y N D | YND | Y N D |
| (Yes/No/Don't Know) | | | | | |
| → If yes, what medication(s)? | | | | | |
| → Please circle those that were provided for you at | | | | | |
| your pre-travel consultation with the study clinic. | | | | | |
| What city(ies) and country(ies) have you been in during the past 24 hours? | | | | | |
| Please write answers to all questions in the corresponding box. | | | | | |
| Trease write union to an question in the corresponding now | | | | | |
| Have you eaten any of the following in the past 24 hours? | | | | | |
| (Yes/No/Don't Know) | | | | | |
| → Fermented or pickled foods (e.g., bean paste, fish | Y N D | Y N D | Y N D | Y N D | Y N D |
| kimchi, etc.) | | | | | |
| → Yogurt | Y N D | Y N D | Y N D | Y N D | Y N D |
| Comments: | | | | | |
| Comments. | | | | | |

| PARTICIPANT UNIQUE ID: |
|------------------------|
| GROUP ID: |

| | Day 16 | Day 17 | Day 18 | Day 19 | Day 20 |
|---|---|---|---|---|---|
| Please write the calendar date that corresponds to each day of your trip. Day 1 is your first day of arrival in the country. | | | | | |
| Number of tablets taken in the morning (maximum 4) | | | | | |
| Number of tablets taken in the afternoon/evening (maximum 4) | | | | | |
| Symptoms in the prior 24 hours (check off all that apply) | | | | | |
| Fever | | | | | |
| Nausea | | | | | |
| Vomiting | | | | | |
| Loose stools (less than three in a 24 hour period) | | | | | |
| Diarrhea (three or more loose stools in 24 hours) | | | | | |
| Bloody diarrhea | | | | | |
| Constipation | | | | | |
| Dark or black stool | | | | | |
| Dark or black tongue | | | | | |
| Abdominal pain | | | | | |
| Abdominal cramps | | | | | |
| Urgency to relieve oneself (in reference to stool) | | | | | |
| Bloating | | | | | |
| Flatulence/gas | | | | | |
| Congestion/runny nose | | | | | |
| Sore throat | | | | | |
| Cough | | | | | |
| Rash | | | | | |
| Headache | | | | | |
| Dizziness | | | | | |
| Ringing in your ears | | | | | |
| Muscle pain/soreness | | | | | |
| Joint pain/swelling/redness | | | | | |
| Drowsiness (severe) | | | | | |
| Confusion | | | | | |
| Denression | П | П | П | П | П |

| Other (list/describe): | | | | | |
|---|---|---|---|---|---|
| other (had describe). | _ | _ | | | |
| Medical care | | | | | |
| Did you seek medical care for one or more of these symptoms? | Y N D | Y N D | Y N D | Y N D | Y N D |
| (Yes/No/Don't Know) | | | | | |
| → If yes, where? (check the corresponding box(es)) | | | | | |
| A doctor's office | | | | | |
| Urgent care clinic (outpatient) | | | | | |
| Emergency room | | | | | |
| Hospital outpatient clinic setting | | | | | |
| Hospital inpatient ward – hospitalized | | | | | |
| Other (specify) | | | | | |
| → Was your diagnosis travelers' diarrhea? | Y N D | Y N D | Y N D | Y N D | Y N D |
| (Yes/No/Don't Know) | | | | | |
| Have you started any medications in the past 24 hours? | Y N D | Y N D | Y N D | YND | Y N D |
| (Yes/No/Don't Know) | | | | | |
| → If yes, what medication(s)? | | | | | |
| → Please circle those that were provided for you at | | | | | |
| your pre-travel consultation with the study clinic. | | | | | |
| What city(ies) and country(ies) have you been in during the past 24 hours? | | | | | |
| Please write answers to all questions in the corresponding box. | | | | | |
| Trease write union to an question in the corresponding now | | | | | |
| Have you eaten any of the following in the past 24 hours? | | | | | |
| (Yes/No/Don't Know) | | | | | |
| → Fermented or pickled foods (e.g., bean paste, fish | Y N D | Y N D | Y N D | Y N D | Y N D |
| kimchi, etc.) | | | | | |
| → Yogurt | Y N D | Y N D | Y N D | Y N D | Y N D |
| Comments: | | | | | |
| Comments. | | | | | |

| PARTICIPANT UNIQUE ID: |
|------------------------|
| GROUP ID: |

| | Day 21 |
|---|---|
| Please write the calendar date that corresponds to each day of your trip. Day 1 is your first day of arrival in the country. | |
| Number of tablets taken in the morning (maximum 4) | |
| Number of tablets taken in the afternoon/evening (maximum 4) | |
| Symptoms in the prior 24 hours (check off all that apply) | • • • |
| Fever | |
| Nausea | |
| Vomiting | |
| Loose stools (less than three in a 24 hour period) | |
| Diarrhea (three or more loose stools in 24 hours) | |
| Bloody diarrhea | |
| Constipation | |
| Dark or black stool | |
| Dark or black tongue | |
| Abdominal pain | |
| Abdominal cramps | |
| Urgency to relieve oneself (in reference to stool) | |
| Bloating | |
| Flatulence/gas | |
| Congestion/runny nose | |
| Sore throat | |
| Cough | |
| Rash | |
| Headache | |
| Dizziness | |
| Ringing in your ears | |
| Muscle pain/soreness | |
| Joint pain/swelling/redness | |

| Drowsiness (severe) | |
|---|---|
| Confusion | |
| Depression | |
| Other (list/describe): | |
| Medical care | |
| Did you seek medical care for one or more of these symptoms? | Y N D |
| (Yes/No/Don't Know) | T IN D |
| → If yes, where? (check the corresponding box(es)) | |
| A doctor's office | • • • • |
| Urgent care clinic (outpatient) | |
| Emergency room | |
| Hospital outpatient clinic setting | |
| Hospital inpatient ward – hospitalized | |
| Other (specify) | |
| → Was your diagnosis travelers' diarrhea? | YND |
| (Yes/No/Don't Know) | TND |
| Have you started any medications in the past 24 hours? | YND |
| (Yes/No/Don't Know) | IND |
| → If yes, what medication(s)? | |
| → Please circle those that were provided for you at | |
| your pre-travel consultation with the study clinic. | |
| What city(ies) and country(ies) have you been in during the past 24 hours? | |
| Please write answers to all questions in the corresponding box. | |
| Have you eaten any of the following in the past 24 hours? | |
| (Yes/No/Don't Know) | |
| → Fermented or pickled foods (e.g., bean paste, fish | YND |
| kimchi, etc.) | |
| → Yogurt | YND |
| Comments: | |



# **Post-travel Questionnaire**

| PARTICIPANT UNIQUE ID: |
|------------------------|
| GROUP ID: |

# 1. Have you had any of the following symptoms since returning home from your trip (circle all that apply)?

| ymptom | Duration (in days) |
|----------------------------------------------------|--------------------|
| Fever | |
| Nausea | |
| Vomiting | |
| Loose stools (less than three in a 24 hour period) | |
| Diarrhea (three or more loose stools in 24 hours) | |
| Bloody diarrhea | |
| Constipation | |
| Dark or black stool | |
| Dark or black tongue | |
| Abdominal pain | |
| Abdominal cramps | |
| Fecal urgency | |
| Bloating | |
| Flatulence/gas | |
| Congestion/runny nose | |
| Sore throat | |
| Cough | |
| Rash | |
| Headache | |
| Dizziness | |
| Ringing in your ears | |
| Muscle pain/soreness | |
| Joint pain/swelling/redness | |
| Drowsiness (severe) | |
| Confusion | |
| Depression | |
| Other (list/describe): | |
| Don't know | |
| I would rather not answer | |

### 2. Did you start taking any of the following medications since you arrived home (circle all that apply)?

- a. Oral or intravenous (IV) antibiotics (e.g., azithromycin [Zithromax], ciprofloxacin [Cipro], rifaximin [Xifaxan], doxycycline or minocycline, metronidazole [Flagyl], cotrimoxazole [Bactrim or Septra], penicillins [e.g., amoxicillin, Augmentin], or cephalosporins [e.g., Keflex])
- **b.** Antidiarrheals (e.g., bismuth subsalicylate [Pepto Bismol/Kaopectate])
- c. Antimotility agents (e.g., loperamide [Imodium])
- d. H2 blocker (e.g., ranitidine [Zantac], cimetidine [Tagamet], famotidine [Pepcid])
- **e. Proton pump inhibitor** (e.g., omeprazole [Prilosec], pantoprazole [Protonix], lansoprazole [Prevacid], esomeprazole [Nexium])
- **f.** Other antacids (e.g., calcium carbonate [Tums/Rolaids], Maalox/Mylanta)
- **g. Probiotics** (Yogurts and other fermented dairy products are probiotics. Probiotics can also take the form of capsules, pills, or powders. Probiotics also include any foods or drinks labeled as containing "live and active cultures" or "probiotics")
- **h.** Oral or intravenous steroids (e.g., prednisone, hydrocortisone)
- i. Local/natural or herbal remedies (herbs, etc.)
- j. Other:

\_\_\_\_\_

3. Did you experience any of the following at any point during your travels?

| Symptom | (Yes/No/Don't Know) | If yes, what was the duration (in days)? |
|---|---|---|
| Ringing in your ears | Y N D | |
| Constipation | Y N D | |
| Dark or black stool | Y N D | |
| Dark or black tongue | Y N D | |
| Drowsiness | Y N D | |
| Nausea | Y N D | |
| Vomiting | Y N D | |
| Rash | Y N D | |
| Other (list/describe): | | |

#### 4. Did you seek medical care for an illness since returning to the United States after your trip?

- a. Yes
- b. No
- c. Don't know
- d. I would rather not answer

#### If yes to question 4, where did you seek and receive care?

- a. A doctor's office
- b. Urgent care clinic (outpatient)
- c. Emergency room
- d. Hospital outpatient clinical setting
- e. Hospital inpatient ward hospitalized
- f. Other (please specify)

\_\_\_\_\_\_

| | • | n 4, were you told that your illness was related to travel? | |
|---|---|---|---|
| | a. Yes | | |
| | b. No | | |
| | c. Don't kn | | |
| | d. I would r | rather not answer | |
| | If yes to question | n 4, were you told that you had travelers' diarrhea? | |
| | a. Yes | | |
| | b. No | | |
| | c. Don't kn | ow | |
| | d. I would r | rather not answer | |
| | If yes to question | n 4, were you told that you had a bacteria that was resistant to | antibiotics? |
| | a. Yes | | |
| | b. No | | |
| | c. Don't kn | ow | |
| | d. I would r | rather not answer | |
| | Did vou travel to | any countries not discussed during your pre-travel visit? | |
| | a. Yes | , any commission and anomaly can produce the state. | |
| | b. No | | |
| | c. Don't kn | ΟW | |
| | | rather not answer | |
| | If yes to question | n 5, please list the new countries you visited, the location(s) vis | ited and the number |
| | of days in each of | | itea, and the number |
| ( | Country name | Specific location(s) to be visited | Number of days in |
| | | (e.g., city/town, attraction) | this country |
| , | | | |

- 6. Did you not travel to a country you discussed at your pre-travel visit?
  - a. Yes

5.

| L- | N | _ |
|----|-----|----|
| r١ | 1/1 | 71 |

- c. Don't know
- d. I would rather not answer

If yes to question 6, please list the countries you did not visit.

| | Country name |
|----|--------------|
| 1. | |
| 2. | |
| 3. | |
| 4. | |
| 5. | |

- 7. Did the time you spent in each country change from what you reported at your pre-travel visit?
  - a. Yes
  - b. No
  - c. Don't know
  - d. I would rather not answer

If yes to question 7, please list the countries in which the amount of time spent changed, including the number of days actually spent in each country:

| Country name | Number of days in this country |
|--------------|--------------------------------|
| 1. | |
| 2. | |
| 3. | |
| 4. | |
| 5. | |

# This survey is now completed.

Thank you very much for your time.

# [PLEASE SEE SEPARATE DOCUMENT]

# APPENDIX G: Follow-up Phone Call Schedule

| | 7 days before travel | 5 days before travel | 3 days before travel | 1 day before<br>travel |
|---|---|---|---|---|
| Review all screening questionnaire answers with the participant, perform the pre-travel questionnaire, and provide a reminder for stool sample submission | X | X | X | X |
| | | 5 L C | - · · · · | 40 1 6 |
| | 3 days after travel | 5 days after travel | 7 days after travel | 10 days after travel |
| Reminder for post-travel questionnaire and stool sample submission | X | Х | х | X |

#### **APPENDIX H: Promotion Materials**

#### Facebook:

Traveling overseas? Our clinic is offering an opportunity to enroll in a study regarding travelers diarrhea. You'll be compensated for your participation. Check out our website at <a href="www.travelhealth.net">www.travelhealth.net</a> for more information!

Traveling abroad? Consider enrolling in our study regarding travelers' diarrhea. Visit our website at <a href="https://www.travelhealth.net">www.travelhealth.net</a> or schedule an appointment by calling 646-374-4132 to learn more!

Participate in our study regarding travelers' diarrhea! If you're interested and have international travel plans, check out our website at <a href="https://www.travelhealth.net">www.travelhealth.net</a> for more information.

### Twitter (@nyctravelmed):

Traveling abroad? Enroll in our study regarding travelers' diarrhea. More info at <a href="www.travelhealth.net">www.travelhealth.net</a>! [102 characters]

Make \$ during travel & help us learn more - enroll in a study regarding travelers' diarrhea. Visit <a href="https://www.travelhealth.net">www.travelhealth.net</a>! [121 characters]

Our clinic is now enrolling for a study regarding travelers' diarrhea. Make \$ and learn more at <a href="https://www.travelhealth.net">www.travelhealth.net</a>! [117 characters]

### Instagram:



[stock image from public health image library]

Participate in a study regarding travelers' diarrhea! Visit our website at <u>www.travelhealth.net</u> for more info on how to participate!



[stock image from public health image library]

Traveling internationally? Participate in a study regarding travelers' diarrhea and receive compensation for your time! Visit our website at <a href="https://www.travelhealth.net">www.travelhealth.net</a> for more info!

Clinic website:

### Participate in a Study to Prevent Travelers' Diarrhea

The New York Travel and Tropical Medicine Clinic is now enrolling international travelers in a study of a medication to prevent travelers' diarrhea. Participants will be compensated for their time. If you or someone you know is 18 or older, is traveling internationally in the upcoming months, and is interested in learning more, give us a call or schedule an appointment with a provider.

Newspaper (Manhattan and/or Brooklyn):

#### Traveling internationally soon?

The New York Travel and Tropical Medicine Clinic is now enrolling international travelers in a study of a medication to prevent travelers' diarrhea. Participants will be compensated for their time! If you or someone you know is 18 or older, is traveling internationally in the upcoming months, and is interested in learning more, give us a call at 646-374-4132 to schedule an appointment. Visit us at <a href="https://www.travelhealth.net">www.travelhealth.net</a>.

# Social media management plan:

- 1. User comments will be monitored for accuracy weekly
- 2. For any technical issues regarding posts on Facebook, Twitter, and Instagram, those platforms will be notified of issues. A web management organization assists with the clinic website.
- 3. Inappropriate or misleading comments will be addressed immediately. Depending on the nature of the comment, it will be addressed in public forum or removed and addressed specifically with the individual who posted the comment.

# APPENDIX I: Data Analysis Table Shells

**Table 1. Baseline Characteristics of Participants** 

| | BSS | Placebo | P-value |
|-----------------------------|-----|---------|---------|
| Demographics | | | |
| Age | | | |
| Sex | | | |
| Race | | | |
| Ethnicity | | | |
| Medical History | | | |
| Chronic medical conditions | | | |
| Tinnitis | | | |
| Antibiotics between 30 to | | | |
| 90 days prior to travel | | | |
| Probiotics within 30 days | | | |
| Travel | | | |
| Duration of travel | | | |
| Primary reason for travel | | | |
| Secondary reasons for | | | |
| travel | | | |
| Exposures during travel | | | |
| Fermented or pickled foods | | | |
| Yogurt | | | |
| Attended provider (by type) | | | |

Table 2. Odds ratios (OR) of TD associated with BSS among international travelers, adjusting for select factors

| | Total,<br>N | TD,<br>% | OR (95% CI) |
|-------------------|-------------|----------|-------------|
| Tablets | | | |
| BSS | | | |
| Placebo | | | Ref |
| Age groups, years | | | |
| ≥18 | | | |
| Sex | | | |
| Male | | | |
| Female | | | Ref |
| Race/ethnicity | | | |
| Travel region | | | |
| Travel duration | | | |

Table 3. The proportion of participants having resistance genes before and after travel; acquiring, losing, or maintaining genes after travel

| | All participants | BSS | Placebo | P-value |
|---------------------|------------------|-----|---------|---------|
| Pre-travel | | | | |
| Gene 1 | | | | |
| Gene 2 | | | | |
| Gene 3 | | | | |
| Gene 4 | | | | |
| Post-travel | | | | |
| Gene 1 | | | | |
| Gene 2 | | | | |
| Gene 3 | | | | |
| Gene 4 | | | | |
| Acquisition of gene | | | | |
| Gene 1 | | | | |
| Gene 2 | | | | |
| Gene 3 | | | | |
| Gene 4 | | | | |
| Loss of gene | | | | |
| Gene 1 | | | | |
| Gene 2 | | | | |
| Gene 3 | | | | |
| Gene 4 | | | | |
| Maintenance of | | | | |
| gene | | | | |
| Gene 1 | | | | |
| Gene 2 | | | | |
| Gene 3 | | | | |
| Gene 4 | | | | |

### APPENDIX J: Auto-Generate Email for Questionnaires

Greetings,

It's time to complete your "Day X" survey!

If your travel plans change or you need to contact us regarding the study, please contact us at: NYTravelStudy@gmail.com.

Thank you,

The New York Center for Travel and Tropical Medicine

You may open the survey in your web browser by clicking the link below:

Bismuth subsalicylate's Role in the Prevention of Travelers' Diarrhea: Daily Questionnaire

If the link above does not work, try copying the link below into your web browser: <a href="https://rdcp.cdc.gov/surveys/?s=QbH5omcTYB">https://rdcp.cdc.gov/surveys/?s=QbH5omcTYB</a>

This link is unique to you and should not be forwarded to others.



Thank you for your participation in this study to see if bismuth subsalicylate (BSS) prevents travelers' diarrhea or prevents you from being colonized with drug-resistant bacteria in your gut.

### **Summary of Procedures for Participants:**

- Approximately 7 days prior to your departure, you will receive a call from clinic personnel. They will verify that the responses you provided to the brief questionnaire at your enrollment visit are still accurate. They will also administer a <a href="Pre-Travel Questionnaire">Pre-Travel Questionnaire</a> over the phone and remind you to submit your first stool sample.
  - After this call, you will receive an email containing your Study ID, Group ID, and a link for you to fill out some addition information about your upcoming trip.
  - ❖ You <u>MUST</u> complete this questionnaire prior to departing for your trip. *If you do not complete it, you will be excluded from the study.*
  - If you do not receive an email within 24 hours of completing the enrollment form, please contact the travel clinic.
  - Stool sample mailing materials will be provided to you at your pre-travel visit. If they were not received or if they were misplaced, please contact the travel clinic.
- ❖ You will receive your first <u>Daily Travel Log</u> via email on your first day of travel in Africa (excluding South Africa) and/or South East or South Central Asia. You will continue to receive these emails daily for the duration of your travels in these regions.
  - Complete the Daily Travel Log after taking your second dose of tablets (e.g., evening).
  - ❖ You will have 48 hours to complete each Daily Travel Log entry. You will receive an email reminder every 12 hours until each questionnaire has been completed or expires.
  - If you have limited internet access or are unable to access the link, please complete the Daily Travel Log on the paper form provided instead.
  - If you are filling out the Daily Travel Log on the paper copies provided and are unable to complete a daily entry within 48 hours, please leave that day blank.
- On the day you return to the US, you will receive an additional email asking you to complete the <u>Post-Travel Questionnaire</u>.
  - ❖ You have 10 days to complete this questionnaire. You will receive an email reminder every 48 hours until the post-travel questionnaire has been completed or expires.
  - You will also need to <u>submit your second stool sample</u> and any paper Travel Log Forms that were completed in lieu of the web-based form. Materials to mail the stool sample and the questionnaires should have been provided to you at your pre-travel visit. If they were not recieved or if they were misplaced, please contact the travel clinic.

If you do not receive an email within 24 hours of returning from your trip, please contact the travel clinic.

If your travel plans change or if you have any questions regarding the study, please contact The New York Center for Travel and Tropical Medicine:

**Phone: +1** (646) 461-1125

E-mail: <u>NYTravelStudy@gmail.com</u>